CLINICAL TRIAL: NCT02408549
Title: An Open-label, Multicenter Extension Study to Evaluate the Long-term Safety and Efficacy of Lacosamide as Adjunctive Therapy for Uncontrolled Primary Generalized Tonic-Clonic Seizures in Subjects With Idiopathic Generalized Epilepsy
Brief Title: Safety and Efficacy of Lacosamide as Additional Therapy in Patients Suffering From Epileptic Tonic-Clonic Seizures
Acronym: VALUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0012; 2012-001770-29 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; Epilepsy; Children; Primary Generalized Tonic Clonic seizures; Idiopathic Generalized Epilepsy; Adults
MeSH Terms: conditions — Epilepsy; Epilepsy, Idiopathic Generalized | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lacosamide (Experimental): Start dose
  SP0982 completers at V1:
  * LCM 10 mg/kg/day for pediatric subjects weighing <30 kg
  * LCM 8 mg/kg/day for pediatric subjects weighing ≥ 30kg to <50 kg
  * LCM 400 mg/day (200 mg bid) for adult subjects (≥18 years of age) or pediatric subjects weighing ≥50 kg
  SP0982 Baseline failures at V1:
  * LCM 2 mg/kg/day for pediatric subjects weighing <50 kg
  * LCM 100 mg/day (50 mg bid) for adult subjects (≥18 years of age) or pediatric subjects weighing ≥50 kg
  Oral solution (pediatric subjects <50 kg):
  * Minimum LCM dose: 4 mg/kg/day
  * Maximum LCM dose: 12 mg/kg/day
  Tablets (pediatric subjects ≥50kg):
  * Minimum LCM dose: 200 mg/day
  * Minimum LCM dose: 600 mg/day
  Tablets (adult subjects):
  * Minimum LCM dose: 200 mg/day
  * Maximum LCM dose: 800 mg/day
  Interventions: Drug: Lacosamide Tablet; Drug: Lacosamide Oral Solution

INTERVENTIONS:
Drug: Lacosamide Tablet — * Active substance: Lacosamide
  * Pharmaceutical form: Tablet
  * Concentration: 50 mg and 100 mg
  * Route of Administration: Oral administration
  Other Names: Vimpat; LCM
Drug: Lacosamide Oral Solution — * Active substance: Lacosamide
  * Pharmaceutical form: Oral solution
  * Concentration: 10 mg/ml
  * Route of Administration: Oral administration
  Other Names: Vimpat; LCM

SUMMARY:
Assessment of long-term safety and efficacy of oral lacosamide (LCM) as an adjunctive therapy for uncontrolled primary generalized tonic-clonic seizures (PGTCS) in subjects >= 4 years of age with idiopathic generalized epilepsy (IGE). This study will enroll subjects from the LCM SP0982 [NCT02408523] study.

ELIGIBILITY:
Inclusion Criteria:

- Subject must have completed or be an eligible Baseline failure from the parent study (SP0982 [NCT02408523]). Note: Other subjects screened for SP0982 may be considered for roll-over to EP0012 if the investigator considers that the subject could benefit from treatment with open-label lacosamide (LCM) and based on prior discussion with and approval from the UCB Study Physician or representative

Exclusion Criteria:

* Subject is receiving any investigational drugs or using any experimental devices in addition to lacosamide (LCM)
* Subject meets the withdrawal criteria for SP0982 or is experiencing an ongoing serious adverse event (SAE)
* Subject has an active suicidal ideation as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Since Last Visit" version of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Subject has >=2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%). For all subjects who entered EP0012 directly with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report form (eCRF). Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit may be repeated once for confirmation.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (87):
- United States (16):
  - EP0012 5, Little Rock, Arkansas
  - EP0012 8, Santa Monica, California
  - Ep0012 31, Colorado Springs, Colorado
  - Ep0012 42, Loxahatchee Groves, Florida
  - Ep0012 13, Panama City, Florida
  - EP0012 2, Port Charlotte, Florida
  - Ep0012 15, Boise, Idaho
  - Ep0012 21, Peoria, Illinois
  - Ep0012 25, Golden Valley, Minnesota
  - Ep0012 43, New York, New York
  - Ep0012 53, Austin, Texas
  - Ep0012 50, Greenville, Texas
  - Ep0012 34, Houston, Texas
  - Ep0012 38, San Antonio, Texas
  - Ep0012 27, Renton, Washington
  - Ep0012 23, Madison, Wisconsin
- Australia (4):
  - Ep0012 980, Chatswood
  - Ep0012 985, Heidelberg
  - Ep0012 986, Melbourne
  - Ep0012 981, Parkville
- Brazil (6):
  - Ep0012 181, Curitiba
  - Ep0012 180, Florianópolis
  - Ep0012 186, Passo Fundo
  - Ep0012 185, Porto Alegre
  - Ep0012 188, Rio de Janeiro
  - Ep0012 183, São Paulo
- Bulgaria (2):
  - Ep0012 500, Blagoevgrad
  - Ep0012 501, Sofia
- China (3):
  - Ep0012 971, Beijing
  - Ep0012 976, Changchun
  - Ep0012 972, Shanghai
- Czechia (4):
  - Ep0012 550, Ostrava- Poruba
  - Ep0012 553, Prague
  - Ep0012 556, Prague
  - Ep0012 552, Zlín
- France (3):
  - Ep0012 255, Bron
  - Ep0012 252, Lille
  - Ep0012 251, Nancy
- Germany (3):
  - Ep0012 303, Erlangen
  - Ep0012 314, Freiburg im Breisgau
  - Ep0012 311, Marburg
- Hungary (2):
  - Ep0012 600, Budapest
  - Ep0012 603, Szeged
- Israel (2):
  - Ep0012 850, Rehovot
  - Ep0012 851, Tel Litwinsky
- Ep0012 351, Torino, Italy
- Japan (11):
  - Ep0012 906, Fukuoka
  - Ep0012 910, Gifu
  - Ep0012 903, Hamamatsu
  - Ep0012 902, Hiroshima
  - Ep0012 912, Kagoshima
  - Ep0012 914, Kodaira
  - Ep0012 909, Kokubunji-shi
  - Ep0012 901, Niigata
  - Ep0012 911, Omura-shi
  - Ep0012 900, Sapporo
  - Ep0012 908, Shinjuku-ku
- Ep0012 161, Guadalajara, Mexico
- Poland (9):
  - Ep0012 657, Częstochowa
  - Ep0012 655, Gdansk
  - Ep0012 652, Gliwice
  - Ep0012 651, Katowice
  - Ep0012 653, Katowice
  - Ep0012 654, Katowice
  - Ep0012 656, Tyniec Mały
  - Ep0012 650, Warsaw
  - Ep0012 659, Warsaw
- Ep0012 451, Lisbon, Portugal
- Romania (2):
  - Ep0012 704, Iași
  - Ep0012 700, Timișoara
- Russia (6):
  - Ep0012 750, Kazan'
  - Ep0012 758, Pyatigorsk
  - Ep0012 755, Saint Petersburg
  - Ep0012 756, Saint Petersburg
  - Ep0012 752, Samara
  - Ep0012 757, Yekaterinburg
- Slovakia (2):
  - Ep0012 821, Bardejov
  - Ep0012 823, Hlohovec
- South Korea (3):
  - Ep0012 940, Daegu
  - Ep0012 941, Seoul
  - Ep0012 944, Seoul
- Spain (4):
  - Ep0012 402, Barcelona
  - Ep0012 406, Córdoba
  - Ep0012 407, Madrid
  - Ep0012 403, Seville
- Taiwan (2):
  - Ep0012 961, Taichung
  - Ep0012 960, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Derived] Vossler DG, Farkas MK, Poverennova I, Watanabe M, Conrath P, Dimova S, McClung C, Roebling R, Williams P, O'Brien TJ; EP0012 Study Group. Long-term safety and efficacy of adjunctive lacosamide in the treatment of generalized onset tonic-clonic seizures: An open-label extension trial. Epilepsia. 2024 Dec;65(12):3488-3500. doi: 10.1111/epi.18158. Epub 2024 Oct 26. PMID 39460685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2015 and concluded in March 2023. Study participants from SP0982 [NCT02408523], who met EP0012 eligibility criteria were enrolled.
Pre-assignment Details: The Participant Flow refers to the Safety Set. The Safety Set included all study participants who received at least 1 dose of Investigational medicinal product (IMP) during this study.
Groups:
- All Participants (Lacosamide): Participants included in this treatment group received at least one dose of LCM as EP0012 protocol entry criteria. The dose range for pediatric participants weighing <50 kg is from 4 mg/kg/day (oral solution) to 12 mg/kg/day (oral solution), for pediatric participants weighing ≥50 kg, the dose range is from 200 mg/day (tablets) to 600 mg/day (tablets) and for adult participants, the dose range is from 200 mg/day to 800mg/day (tablets) during the Treatment Period. The LCM dose may be increased or decreased at the investigator's discretion after the study participant received the first dose of LCM in the study. Pediatric participants who initially started on oral solution might have transferred to tablets at Investigator's discretion after achieving >=50 kgs. LCM was administered orally, twice daily (bid), up to approximately 5 years. Treatment was continued for at least 2 years for adult participants and up to approximately 5 years for pediatric participants.
Period: Overall Study
Arm/Group | All Participants (Lacosamide)
Started | 239
Completed | 157
Not Completed | 82
Not completed — Adverse Event | 15
Not completed — Death | 4
Not completed — Lack of Efficacy | 17
Not completed — Protocol Violation | 4
Not completed — Lost to Follow-up | 6
Not completed — Consent withdrawn | 30
Not completed — Neurology research program closing at site | 1
Not completed — Site closure | 1
Not completed — Pregnancy | 1
Not completed — Withdrawal of consent due to business trip | 1
Not completed — Subject moved to another place, far from site | 1
Not completed — Study terminated at site | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all study participants who received at least 1 dose of IMP during this study.
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (12.6)
Age, Customized [Count of Participants; unit: Participants]
  ≥4-<12 years | 16
  12-<18 years | 28
  18-<65 years | 194
  ≥65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1
  Asian | 48
  Black | 4
  White | 178
  Other/Mixed | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 211

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants With Treatment-emergent Adverse Events (TEAEs) Over the Duration of the Treatment Period
Description: AEs were considered treatment-emergent if event had onset on or after date of first study medication dose in EP0012 and within 30 days following last study medication dose or events whose intensity worsened on or after date of first study medication dose and within 30 days following date of last study medication administration. Adverse Events were reported spontaneously by the participant and/or caregiver or observed by the investigator.
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
Participants | 222

2. Primary Outcome: Number of Study Participants Withdrawn Due to TEAEs
Description: as for outcome 1
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
Participants | 19

3. Primary Outcome: Number of Study Participants With New Appearance of Absence and/or Myoclonic Seizures During the Treatment Period
Description: The number of study participants with appearance of new absence and/or myoclonic seizure types experienced during the Treatment Period but who did not experience in Combined Baseline Period or in seizure classification history, before taking LCM were reported. To determine appearance of new seizure type, the Combined Baseline Period was used. Thus, the participants who directly enrolled into EP0012, the Baseline absence, and/or myoclonic seizure data from SP0982's 4-week Prospective Baseline Period were combined with any reported Baseline absence, and myoclonic seizure information in the daily seizure diary from EP0012 (reported before first dose in EP0012) to recalculate the study participant's Baseline variables such as days with absence, and/or myoclonic seizures per 28 days.
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
Participants
  Absence seizures | 3
  Myoclonic seizures | 5

4. Primary Outcome: Number of Study Participants With an Increase of up to 25% in Days With Absence Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of up to 25% in the number of days with absence seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with absence seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years), compared to the Prospective SP0982 Baseline Period
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Here, Number of participants analyzed included those participants who were evaluable for the assessment (absence seizures).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 93
Participants | 5

5. Primary Outcome: Number of Study Participants With an Increase of Greater Than (>)25% to 50% in Days With Absence Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of >25% to 50% in the number of days with absence seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with absence seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 93
Participants | 1

6. Primary Outcome: Number of Study Participants With an Increase of >50% to 75% in Days With Absence Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of >50% to 75% in the number of days with absence seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with absence seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 93
Participants | 0

7. Primary Outcome: Number of Study Participants With an Increase of >75% in Days With Absence Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of >75% in the number of days with absence seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with absence seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 93
Participants | 0

8. Primary Outcome: Number of Study Participants With an Increase of up to 25% in Days With Myoclonic Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of up to 25% in the number of days with myoclonic seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with myoclonic seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Here, Number of participants analyzed included those participants who were evaluable for the assessment (myoclonic seizures).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 96
Participants | 4

9. Primary Outcome: Number of Study Participants With an Increase of >25% to 50% in Days With Myoclonic Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of >25% to 50% in the number of days with myoclonic seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with myoclonic seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 96
Participants | 1

10. Primary Outcome: Number of Study Participants With an Increase of >50% to 75% in Days With Myoclonic Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of >50% to 75% in the number of days with myoclonic seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with myoclonic seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 96
Participants | 1

11. Primary Outcome: Number of Study Participants With an Increase of >75% in Days With Myoclonic Seizures Per 28 Days During the Treatment Period as Compared to the Prospective Baseline (of Study SP0982)
Description: The number of participants experiencing an increase of >75% in the number of days with myoclonic seizures per 28 days during the Treatment Period compared to the Prospective Baseline Period (for those participants with myoclonic seizure data reported in the 4-week Prospective Baseline Period in SP0982) were reported. This period started on the day of Visit 1 of SP0982 and ended the day before Visit 2 of SP0982. For the direct enrollers into EP0012, Prospective Baseline ended the day before Visit 1 (or prior to first dose) of EP0012.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 96
Participants | 2

12. Primary Outcome: Percentage of Study Participants With at Least 50% Worsening in Days With Absence Seizures
Description: Seizure worsening was defined as a participant experiencing >=50% increase in the number of days with absence seizures per 28 days from Prospective Baseline. Percentages for seizure worsening were based on those participants who have reported a history of or an occurrence of absence seizures in Prospective Baseline or the Treatment Period.
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 92
percentage of participants | 0

13. Primary Outcome: Percentage of Study Participants With at Least 50% Worsening in Days With Myoclonic Seizures
Description: Seizure worsening was defined as a participant experiencing >=50% increase in the number of days with myoclonic seizures per 28 days from Prospective Baseline. Percentages for seizure worsening were based on those participants who have reported a history of or an occurrence of myoclonic seizures in Prospective Baseline or the Treatment Period.
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 95
percentage of participants | 3.2

14. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Hemoglobin)
Description: TEMA values are defined in the Statistical Analysis Plan (SAP) as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Hematology parameter, Hemoglobin were those that were observed post-Baseline (BL) during the Treatment Period but not present at Baseline. For the age range, '2 years (y) to <17 years', the abnormality criteria were '<=95' grams/deciliter (g/dL) (Low) and '>160' g/dL (High). For age range, '>=17 years', the abnormality Criteria were '<=85% of lower limit of normal (LLN)' value (Low) and '>=115% of upper limit of normal (ULN)' value (High) of Hemoglobin in blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Hematology parameter (Hemoglobin) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Low: Week (Wk) 78 (2-<17 y): number analyzed (Participants) | 7
  Low: Week (Wk) 78 (2-<17 y) | 14.3
  Low: Wk 0 (>=17 y): number analyzed (Participants) | 27
  Low: Wk 0 (>=17 y) | 3.7
  Low: Wk 2 (>=17 y): number analyzed (Participants) | 195
  Low: Wk 2 (>=17 y) | 0.5
  Low: Wk 118 (>=17 y): number analyzed (Participants) | 123
  Low: Wk 118 (>=17 y) | 0.8
  Low: Wk 166 (>=17 y): number analyzed (Participants) | 81
  Low: Wk 166 (>=17 y) | 1.2
  Low: Wk 214 (>=17 y): number analyzed (Participants) | 40
  Low: Wk 214 (>=17 y) | 2.5
  Low: Termination Visit (TV) (>=17 y): number analyzed (Participants) | 123
  Low: Termination Visit (TV) (>=17 y) | 1.6

15. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Hematocrit)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Hematocrit were those that were observed post-BL during the Treatment Period but not present at BL. For the age range, '2 years to <17 years', the abnormality criteria were '<=29%' (Low) and '>47%' (High) hematocrit values. For age range, '>=17 years', the abnormality criteria were '<=85% of LLN' (Low) and '>=115% of ULN' (High) of Hematocrit values in blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Hematology parameter (Hematocrit) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  High: Wk 22 (2-<17 y): number analyzed (Participants) | 29
  High: Wk 22 (2-<17 y) | 6.9
  High: Wk 46 (2-<17 y): number analyzed (Participants) | 27
  High: Wk 46 (2-<17 y) | 3.7
  Low: Wk 46 (>=17 y): number analyzed (Participants) | 170
  Low: Wk 46 (>=17 y) | 1.2
  Low: Wk 118 (>=17 y): number analyzed (Participants) | 123
  Low: Wk 118 (>=17 y) | 1.6
  Low: Wk 166 (>=17 y): number analyzed (Participants) | 81
  Low: Wk 166 (>=17 y) | 1.2
  Low: TV (>=17 y): number analyzed (Participants) | 123
  Low: TV (>=17 y) | 0.8

16. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Platelets)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Platelet count were those that were observed post-BL during the Treatment Period but not present at BL. For the age range of '>1 month', the abnormality criteria were '<=100' 10^9/L and '>=600' 10^9/L of Platelets count value.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (platelets) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

17. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Erythrocytes)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Erythrocytes parameter were those that were observed post-BL during the Treatment Period but not present at BL. For the age range, '>=2years', the abnormality criteria were '<3.5' 10^12/L of Erythrocytes value in blood. Early Termination Visit (TV) was last visit in the study (up to approximately 5 years).
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Data for visit (Early TV) wherein at least 1 TEMA value of Hematology parameter (Erythrocytes) observed during the study was reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 59
percentage of participants | 1.7

18. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Leukocytes)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Leukocytes were those that were observed post-BL during the Treatment Period but not present at BL. For all age ranges, the abnormality criteria were '<=3.0' 10^9/L (Low) and '>= 16.0' 10^9/L (High) of Leukocytes values in blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Data for visit (Week 62-Low) wherein at least 1 TEMA value of Hematology parameter (Leukocytes) observed during the study was reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 191
percentage of participants | 0.5

19. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Basophils Absolute)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Basophils Absolute were those that were observed post-BL during the Treatment Period but not present at BL. For the age range, '>1 month', the abnormality criteria were '>=0.4' 10^9/L of Basophils in blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Data for visit (Week 2) wherein at least 1 TEMA value of Hematology parameter (Basophils Absolute) observed during the study was reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 228
percentage of participants | 0.4

20. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Eosinophils Absolute)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Eosinophils Absolute were those that were observed post-BL during the Treatment Period but not present at BL. For the age range, '>1 month', the abnormality criteria were '>=1.0' 10^9/L of Eosinophils in the blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Hematology parameter (Eosinophils Absolute) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 228
percentage of participants
  >=1.0: Wk 2 (>1 month) | 0.9
  >=1.0: Wk 22 (>1 month): number analyzed (Participants) | 215
  >=1.0: Wk 22 (>1 month) | 0.5
  >=1.0: TV (>1 month): number analyzed (Participants) | 134
  >=1.0: TV (>1 month) | 1.5

21. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Lymphocytes Absolute)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Lymphocytes Absolute were those that were observed post-Baseline (BL) during the Treatment Period but not present at Baseline. For the age range, '2 years - <6 years', the abnormality criteria were '<0.7' 10^9/L (Low) and '>6.9' 10^9/L (High). For age range, '>=6 years', the abnormality criteria were '<0.6' 10^9/L (Low) and '>5.0' 10^9/L (High) for Lymphocytes Absolute in the blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Hematology parameter (Lymphocytes Absolute) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 226
percentage of participants
  High: Wk 2 (>=6 y) | 0.4
  High: Wk 78 (>=6 y): number analyzed (Participants) | 63
  High: Wk 78 (>=6 y) | 3.2
  High: Wk 118 (>=6 y): number analyzed (Participants) | 141
  High: Wk 118 (>=6 y) | 0.7

22. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Monocytes Absolute )
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Monocytes Absolute were those that are observed post-BL during the Treatment Period but not present at BL. For the age range, '>1 month', the abnormality criteria was '>=2.0' 10^9/L of Monocytes in blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Monocytes Absolute) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

23. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Hematology Parameters (Neutrophils Absolute)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Neutrophils Absolute were those that were observed post-BL during the Treatment Period but not present at BL. For the age range, '>1 month', the abnormality criteria was '<1.5' 10^9/L of Neutrophils in blood.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Hematology parameter (Neutrophils Absolute) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 228
percentage of participants
  <1.5: Wk 2 (>1 m) | 0.9
  <1.5: Wk 22 (>1 m): number analyzed (Participants) | 215
  <1.5: Wk 22 (>1 m) | 0.5
  <1.5: Wk 46 (>1 m): number analyzed (Participants) | 196
  <1.5: Wk 46 (>1 m) | 0.5
  <1.5: Wk 62 (>1 m): number analyzed (Participants) | 191
  <1.5: Wk 62 (>1 m) | 0.5
  <1.5: Wk 94 (>1 m): number analyzed (Participants) | 162
  <1.5: Wk 94 (>1 m) | 0.6
  <1.5: Wk 214 (>1 m): number analyzed (Participants) | 42
  <1.5: Wk 214 (>1 m) | 2.4

24. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Calcium)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Calcium were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1 year -<17 years', the abnormality criteria were '<=1.85' millimoles per litre (mmol/L) and '>=2.95' mmol/L. For age range, '>=17 years', the abnormality criteria was '<=1.9 mmol/L' and '>=2.75 mmol/L' of serum Calcium.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Calcium) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

25. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Sodium)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Sodium were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>1 month', the abnormality criteria were '<127' mmol/L (Low) and '>151' mmol/L (High) of serum Sodium.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Sodium) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

26. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Potassium)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Potassium were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>=1 year', the abnormality criteria were '<= 3.0' mmol/L (Low) and '>= 6.0' mmol/L (High) of serum Potassium.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Data for visit (Week 2-High) wherein at least 1 TEMA value of Serum chemistry parameter (Potassium) observed during the study was reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 230
percentage of participants | 0.4

27. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Chloride)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Chloride were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>1 month', the abnormality criteria were '<=90' mmol/L (Low) and '>=112' mmol/L (High) of serum Chloride.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (Chloride) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 234
percentage of participants
  High: Wk 2 (>1 m) | 1.3
  High: Wk 22 (>1 m): number analyzed (Participants) | 218
  High: Wk 22 (>1 m) | 2.3
  High: Wk 46 (>1 m): number analyzed (Participants) | 198
  High: Wk 46 (>1 m) | 2.5
  High: Wk 62 (>1 m): number analyzed (Participants) | 194
  High: Wk 62 (>1 m) | 1.5
  High: Wk 78 (>1 m): number analyzed (Participants) | 65
  High: Wk 78 (>1 m) | 3.1
  High: Wk 94 (>1 m): number analyzed (Participants) | 165
  High: Wk 94 (>1 m) | 1.2
  High: Wk 118 (>1 m): number analyzed (Participants) | 145
  High: Wk 118 (>1 m) | 3.4
  High: Wk 214 (>1 m): number analyzed (Participants) | 43
  High: Wk 214 (>1 m) | 2.3
  High: TV (>1 m): number analyzed (Participants) | 145
  High: TV (>1 m) | 1.4

28. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Bicarbonate)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Bicarbonate were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>1 month-<17 years', the abnormality criteria were '<15' mmol/L (Low) and '>38' mmol/L (High). For age range, '>=17 years', the abnormality criteria were '<18' mmol/L (Low) and '>38' mmol/L (High) of serum Bicarbonate.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (Bicarbonate) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 180
percentage of participants
  Low: Wk 2 (>=17 y) | 1.1
  Low: Wk 46 (>=17 y): number analyzed (Participants) | 161
  Low: Wk 46 (>=17 y) | 1.2
  Low: Wk 62 (>=17 y): number analyzed (Participants) | 158
  Low: Wk 62 (>=17 y) | 1.3
  Low: Wk 94 (>=17 y): number analyzed (Participants) | 136
  Low: Wk 94 (>=17 y) | 0.7

29. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Creatinine)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Creatinine were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1-<10 years', the abnormality criteria were '>106.8' micromole per litre (umol/L), for '10-<16 years', the abnormality criteria were '>159.12' umol/L and for '>=16 years', the abnormality criteria was '>=176.8' umol/L for serum Creatinine.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Creatinine) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

30. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Aspartate Aminotransferase)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Aspartate Aminotransferase (AST) were those that were observed post- BL during the Treatment Period but not present at Baseline. For all ages, the abnormality criteria were specified as '≥3.0 units per litre (U/L) x ULN' (High A), '≥5.0 U/L x ULN' (High B), and '≥10.0 U/L x ULN' (High C) of serum AST.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (AST) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  High A: All ages (Early TV): number analyzed (Participants) | 58
  High A: All ages (Early TV) | 1.7
  High A: All ages (TV): number analyzed (Participants) | 144
  High A: All ages (TV) | 0.7
  High B: All ages (TV): number analyzed (Participants) | 144
  High B: All ages (TV) | 0.7
  High C: All ages (TV): number analyzed (Participants) | 144
  High C: All ages (TV) | 0.7

31. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Alanine Aminotransferase)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Alanine Aminotransferase (ALT) were those that were observed post- BL during the Treatment Period but not present at Baseline. For all ages, the abnormality criteria were specified as '≥3.0 U/L x ULN' (High A), '≥5.0 U/L x ULN' (High B), and '≥10.0 U/L x ULN' (High C) of serum ALT.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (ALT) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 234
percentage of participants
  High A: All ages (Wk 2) | 0.4
  High A: All ages (Wk 46): number analyzed (Participants) | 198
  High A: All ages (Wk 46) | 0.5
  High A: All ages (Wk 62): number analyzed (Participants) | 192
  High A: All ages (Wk 62) | 0.5
  High A: All ages (Wk 118): number analyzed (Participants) | 144
  High A: All ages (Wk 118) | 0.7
  High A: All ages (TV): number analyzed (Participants) | 144
  High A: All ages (TV) | 0.7
  High B: All ages (Wk 2) | 0.4

32. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Chemistry Parameters (Total Bilirubin)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Total Bilirubin were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>1 month', the abnormality criteria was '≥34.208' umol/L of serum Bilirubin.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Data for visit (Week 22) wherein at least 1 TEMA value of serum chemistry parameter (Total Bilirubin) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 218
percentage of participants | 0.5

33. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Alkaline Phosphatase)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Alkaline Phosphatase were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '4 years -<10 years', the abnormality criteria was '>=834 U/L', for '10 years -<17 years', the abnormality criteria was '>=1761 U/L' and for '>=17 years', the abnormality criteria was '>=3.0 U/L x ULN' of serum alkaline phosphatase.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Alkaline Phosphatase) with markedly abnormal criteria specified at any visit .
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

34. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Gamma Glutamyl Transferase)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Gamma Glutamyl Transferase (GGT) were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1 year-<13 years', the abnormality criteria was '>=66' U/L (High A), for '13 years-<17 years', the abnormality criteria was '>=126' U/L (High B) and for '>=17 years', the abnormality criteria was '>=3.0 U/L x ULN' (High C) of serum GGT.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (GGT) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  High A: TV (1-<13 y): number analyzed (Participants) | 6
  High A: TV (1-<13 y) | 16.7
  High C: Wk 2 (>=17 y): number analyzed (Participants) | 198
  High C: Wk 2 (>=17 y) | 1.0
  High C: Wk 22 (>=17 y): number analyzed (Participants) | 189
  High C: Wk 22 (>=17 y) | 0.5
  High C: Wk 62 (>=17 y): number analyzed (Participants) | 169
  High C: Wk 62 (>=17 y) | 1.8
  High C: Wk 78 (>=17 y): number analyzed (Participants) | 58
  High C: Wk 78 (>=17 y) | 3.4
  High C: Wk 118 (>=17 y): number analyzed (Participants) | 125
  High C: Wk 118 (>=17 y) | 0.8
  High C: Wk 166 (>=17 y): number analyzed (Participants) | 89
  High C: Wk 166 (>=17 y) | 1.1
  High C:TV (>=17 y): number analyzed (Participants) | 132
  High C:TV (>=17 y) | 0.8

35. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Glucose)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Glucose were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>1 month-<17 years', the abnormality criteria were from '<2.775' mmol/L (Low) and '>=9.99' mmol/L (High). For age range, '>=17 years', the abnormality criteria were '<2.775' mmol/L (Low) and '>=11.1' mmol/L (High) of serum Glucose.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (Glucose) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 195
percentage of participants
  Low: Wk 2 (>=17 y) | 0.5
  Low: Wk 62 (>=17 y): number analyzed (Participants) | 168
  Low: Wk 62 (>=17 y) | 0.6
  Low: Wk 94 (>=17 y): number analyzed (Participants) | 143
  Low: Wk 94 (>=17 y) | 0.7
  Low: Wk 118 (>=17 y): number analyzed (Participants) | 123
  Low: Wk 118 (>=17 y) | 0.8
  High: Wk 2 (>=17 y) | 1.0
  High: Wk 22 (>=17 y): number analyzed (Participants) | 186
  High: Wk 22 (>=17 y) | 1.1
  High: Wk 46 (>=17 y): number analyzed (Participants) | 166
  High: Wk 46 (>=17 y) | 1.2
  High: Wk 62 (>=17 y): number analyzed (Participants) | 168
  High: Wk 62 (>=17 y) | 1.8
  High: Wk 78 (>=17 y): number analyzed (Participants) | 58
  High: Wk 78 (>=17 y) | 3.4
  High: Wk 94 (>=17 y): number analyzed (Participants) | 143
  High: Wk 94 (>=17 y) | 0.7
  High: Wk 118 (>=17 y): number analyzed (Participants) | 123
  High: Wk 118 (>=17 y) | 0.8
  High: Early TV (>=17 y): number analyzed (Participants) | 52
  High: Early TV (>=17 y) | 1.9

36. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Albumin)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Albumin were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '>=1 year to <17 years', the abnormality criteria were '<24' g/L and '>84' g/L and for age range, '>=17 years', the abnormality criteria was '<26' g/L of serum albumin.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Albumin) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

37. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Total Protein)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Total Protein were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1 year to <17 years', the abnormality criteria were '<43' g/L and '>120' g/L. For age range, '>=17 years', the abnormality criteria were '<43' g/L and '>130' g/L of serum protein.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. No participant had TEMA value (Total Protein) with markedly abnormal criteria specified at any visit.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants | 0

38. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Serum Chemistry Parameters (Phosphate)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA laboratory results of Phosphate were those that are observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1 year-<17 years', the abnormality criteria were from '<0.5814' mmol/L (Low) and '>2.3902' mmol/L (High). For age range, '>=17 years', the abnormality Criteria were '<=0.646' mmol/L (Low) and '>=1.938' mmol/L (High) of serum phosphate.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of serum chemistry parameter (Phosphate) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 141
percentage of participants
  Low: Wk 94 (>=17 y) | 0.7
  Low: Wk 118 (>=17 y): number analyzed (Participants) | 123
  Low: Wk 118 (>=17 y) | 0.8

39. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in 12-lead Electrocardiogram (ECG) Parameter (QT Interval)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA ECG results of QT interval parameter were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1 month (m)-<12 years', the abnormality criteria were '>=500 milliseconds (ms)' (Abnormal (Abn) A). For age range, '>=12 years', the abnormality criteria were '>=500 ms' (Abn B) or '>=60 ms increase from Baseline' (Abn C). The abnormality in QT interval was observed at Week 0 as the participant was rolled over from SP0982 study and was constantly having abnormal ECG parameters while in SP0982 and EP0012.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of ECG parameter (QT interval) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 216
percentage of participants
  Abn C: Wk 0 (>=12 years): number analyzed (Participants) | 3
  Abn C: Wk 0 (>=12 years) | 33.3
  Abn C: Wk 2 (>=12 years) | 0.5
  Abn C: Wk 14 (>=12 years): number analyzed (Participants) | 209
  Abn C: Wk 14 (>=12 years) | 3.3
  Abn C: Wk 30 (>=12 years): number analyzed (Participants) | 130
  Abn C: Wk 30 (>=12 years) | 0.8
  Abn B: Wk 46 (>=12 years): number analyzed (Participants) | 188
  Abn B: Wk 46 (>=12 years) | 0.5
  Abn C: Wk 46 (>=12 years): number analyzed (Participants) | 188
  Abn C: Wk 46 (>=12 years) | 2.7
  Abn C: Wk 62 (>=12 years): number analyzed (Participants) | 186
  Abn C: Wk 62 (>=12 years) | 2.2
  Abn C: Wk 78 (>=12 years): number analyzed (Participants) | 61
  Abn C: Wk 78 (>=12 years) | 1.6
  Abn C: Wk 94 (>=12 years): number analyzed (Participants) | 162
  Abn C: Wk 94 (>=12 years) | 2.5
  Abn C: Wk 118 (>=12 years): number analyzed (Participants) | 23
  Abn C: Wk 118 (>=12 years) | 13.0
  Abn C: Wk 142 (>=12 years): number analyzed (Participants) | 58
  Abn C: Wk 142 (>=12 years) | 6.9
  Abn C: Wk 190 (>=12 years): number analyzed (Participants) | 31
  Abn C: Wk 190 (>=12 years) | 3.2
  Abn C: Early TV (>=12 years): number analyzed (Participants) | 52
  Abn C: Early TV (>=12 years) | 3.8
  Abn C: TV (>=12 years): number analyzed (Participants) | 43
  Abn C: TV (>=12 years) | 2.3

40. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in 12-lead ECG Parameter (QTc(F) Interval)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA ECG results of QTc(F) interval were those that are observed post- BL during the Treatment Period but not present at Baseline. For the age range '3 years -<12 years' and '>=12 years- <17 years', the abnormality criteria were from '>440 ms' (Abn A) and '>15% increase from Baseline' value (Abn B). For age range, '>=17 years', the abnormality Criteria were '>450 ms' (Abn C), '>480 ms' (Abn D), '>500 ms' (Abn E) or '>=60 ms increase from Baseline' value (Abn F). The abnormality in QTc(F) interval was observed at Week 0 as the participant was rolled over from SP0982 study and was constantly having abnormal ECG parameters while in SP0982 and EP0012.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of ECG parameter (QTc(F) interval) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Abn C: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn C: Wk 0 (>=17 y) | 33.3
  Abn D: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn D: Wk 0 (>=17 y) | 33.3
  Abn F: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn F: Wk 0 (>=17 y) | 33.3
  Abn C: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn C: Wk 2 (>=17 y) | 1.5
  Abn F: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn F: Wk 2 (>=17 y) | 1.0
  Abn A: Wk 14 (>=12 y-<17 y): number analyzed (Participants) | 18
  Abn A: Wk 14 (>=12 y-<17 y) | 5.6
  Abn C: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn C: Wk 14 (>=17 y) | 2.1
  Abn D: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn D: Wk 14 (>=17 y) | 1.0
  Abn E: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn E: Wk 14 (>=17 y) | 0.5
  Abn F: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn F: Wk 14 (>=17 y) | 3.7
  Abn F: Wk 30 (>=17 y): number analyzed (Participants) | 118
  Abn F: Wk 30 (>=17 y) | 1.7
  Abn C: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn C: Wk 46 (>=17 y) | 5.2
  Abn D: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn D: Wk 46 (>=17 y) | 1.7
  Abn E: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn E: Wk 46 (>=17 y) | 1.2
  Abn F: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn F: Wk 46 (>=17 y) | 2.3
  Abn A: Wk 62 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn A: Wk 62 (>=12 y-<17 y) | 6.3
  Abn B: Wk 62 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn B: Wk 62 (>=12 y-<17 y) | 6.3
  Abn C: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn C: Wk 62 (>=17 y) | 2.4
  Abn D: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn D: Wk 62 (>=17 y) | 0.6
  Abn F: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn F: Wk 62 (>=17 y) | 1.8
  Abn F: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn F: Wk 78 (>=17 y) | 1.8
  Abn C: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn C: Wk 94 (>=17 y) | 2.7
  Abn D: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn D: Wk 94 (>=17 y) | 2.0
  Abn E: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn E: Wk 94 (>=17 y) | 2.0
  Abn F: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn F: Wk 94 (>=17 y) | 3.4
  Abn C: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn C: Wk 118 (>=17 y) | 9.5
  Abn F: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn F: Wk 118 (>=17 y) | 4.8
  Abn C: Wk 142 (>=17 y): number analyzed (Participants) | 47
  Abn C: Wk 142 (>=17 y) | 2.1
  Abn F: Wk 142 (>=17 y): number analyzed (Participants) | 47
  Abn F: Wk 142 (>=17 y) | 2.1
  Abn C: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn C: Early TV (>=17 y) | 6.1
  Abn D: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn D: Early TV (>=17 y) | 2.0
  Abn E: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn E: Early TV (>=17 y) | 2.0
  Abn F: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn F: Early TV (>=17 y) | 4.1
  Abn C: TV (>=17 y): number analyzed (Participants) | 36
  Abn C: TV (>=17 y) | 2.8
  Abn F: TV (>=17 y): number analyzed (Participants) | 36
  Abn F: TV (>=17 y) | 5.6

41. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in 12-lead ECG Parameter (QTc(B) Interval)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA ECG results of QTc(B) interval were those that are observed post- BL during the Treatment Period but not present at Baseline. For the age range '3 years -<12 years' and '>=12 years- <17 years', the abnormality criteria were '>450 ms' (Abn A) and '>15% increase from Baseline' value (Abn B). For age range, '>=17 years', the abnormality criteria were '>450 ms' (Abn C), '>480 ms' (Abn D), '>500 ms' (Abn E) or '>=60 ms increase from Baseline' value (Abn F). The abnormality in QTc(B) interval was observed at Week 0 as the participant was rolled over from SP0982 study and was constantly having abnormal ECG parameters while in SP0982 and EP0012.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of ECG parameter (QTc(B) interval) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Abn C: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn C: Wk 0 (>=17 y) | 33.3
  Abn D: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn D: Wk 0 (>=17 y) | 33.3
  Abn E: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn E: Wk 0 (>=17 y) | 33.3
  Abn F: Wk 0 (>=17 y): number analyzed (Participants) | 3
  Abn F: Wk 0 (>=17 y) | 33.3
  Abn C: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn C: Wk 2 (>=17 y) | 3.6
  Abn F: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn F: Wk 2 (>=17 y) | 2.0
  Abn A: Wk 14 (>=12 y-<17 y): number analyzed (Participants) | 18
  Abn A: Wk 14 (>=12 y-<17 y) | 5.6
  Abn C: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn C: Wk 14 (>=17 y) | 5.8
  Abn D: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn D: Wk 14 (>=17 y) | 1.6
  Abn E: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn E: Wk 14 (>=17 y) | 1.0
  Abn F: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn F: Wk 14 (>=17 y) | 3.7
  Abn C: Wk 30 (>=17 y): number analyzed (Participants) | 118
  Abn C: Wk 30 (>=17 y) | 2.5
  Abn F: Wk 30 (>=17 y): number analyzed (Participants) | 118
  Abn F: Wk 30 (>=17 y) | 1.7
  Abn C: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn C: Wk 46 (>=17 y) | 7.0
  Abn D: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn D: Wk 46 (>=17 y) | 2.9
  Abn E: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn E: Wk 46 (>=17 y) | 1.2
  Abn F: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn F: Wk 46 (>=17 y) | 3.5
  Abn A: Wk 62 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn A: Wk 62 (>=12 y-<17 y) | 6.3
  Abn B: Wk 62 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn B: Wk 62 (>=12 y-<17 y) | 6.3
  Abn C: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn C: Wk 62 (>=17 y) | 2.4
  Abn D: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn D: Wk 62 (>=17 y) | 0.6
  Abn E: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn E: Wk 62 (>=17 y) | 0.6
  Abn F: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn F: Wk 62 (>=17 y) | 3.5
  Abn C: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn C: Wk 78 (>=17 y) | 5.4
  Abn F: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn F: Wk 78 (>=17 y) | 1.8
  Abn C: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn C: Wk 94 (>=17 y) | 5.4
  Abn D: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn D: Wk 94 (>=17 y) | 2.0
  Abn E: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn E: Wk 94 (>=17 y) | 2.0
  Abn F: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn F: Wk 94 (>=17 y) | 3.4
  Abn A: Wk 118 (>=12 y-<17 y): number analyzed (Participants) | 2
  Abn A: Wk 118 (>=12 y-<17 y) | 50.0
  Abn C: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn C: Wk 118 (>=17 y) | 14.3
  Abn D: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn D: Wk 118 (>=17 y) | 4.8
  Abn E: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn E: Wk 118 (>=17 y) | 4.8
  Abn F: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn F: Wk 118 (>=17 y) | 9.5
  Abn A: Wk 142 (>=12 y-<17 y): number analyzed (Participants) | 11
  Abn A: Wk 142 (>=12 y-<17 y) | 9.1
  Abn C: Wk 142 (>=17 y): number analyzed (Participants) | 47
  Abn C: Wk 142 (>=17 y) | 8.5
  Abn F: Wk 142 (>=17 y): number analyzed (Participants) | 47
  Abn F: Wk 142 (>=17 y) | 4.3
  Abn F: Wk 166 (>=17 y): number analyzed (Participants) | 3
  Abn F: Wk 166 (>=17 y) | 33.3
  Abn C: Wk 190 (>=17 y): number analyzed (Participants) | 26
  Abn C: Wk 190 (>=17 y) | 7.7
  Abn F: Wk 190 (>=17 y): number analyzed (Participants) | 26
  Abn F: Wk 190 (>=17 y) | 3.8
  Abn C: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn C: Early TV (>=17 y) | 6.1
  Abn D: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn D: Early TV (>=17 y) | 2.0
  Abn E: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn E: Early TV (>=17 y) | 2.0
  Abn F: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn F: Early TV (>=17 y) | 6.1
  Abn C: TV (>=17 y): number analyzed (Participants) | 36
  Abn C: TV (>=17 y) | 2.8
  Abn D: TV (>=17 y): number analyzed (Participants) | 36
  Abn D: TV (>=17 y) | 2.8
  Abn F: TV (>=17 y): number analyzed (Participants) | 36
  Abn F: TV (>=17 y) | 5.6

42. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in 12-lead ECG Parameter (PR Interval)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA ECG results of PR interval were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '3 years -<12 years', the abnormality criteria were '>180 ms' (Abn A) and '>25% increase from Baseline' value (Abn B). For the age range, '>=12 years - <17 years', the abnormality criteria were '>200 ms' (Abn C) and '>25% increase from Baseline' value (Abn D). For age range, '>=17 years', the abnormality criteria were treatment-emergent values above '>200 ms' (Abn E), '>220 ms' (Abn F), or '>250 ms' (Abn G).
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of ECG parameter (PR interval) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Abn B: Wk 2 (3 y-<12 y): number analyzed (Participants) | 16
  Abn B: Wk 2 (3 y-<12 y) | 6.3
  Abn D: Wk 2 (>=12 y-<17 y): number analyzed (Participants) | 20
  Abn D: Wk 2 (>=12 y-<17 y) | 5.0
  Abn E: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn E: Wk 2 (>=17 y) | 1.5
  Abn F: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn F: Wk 2 (>=17 y) | 0.5
  Abn E: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn E: Wk 14 (>=17 y) | 1.0
  Abn E: Wk 30 (>=17 y): number analyzed (Participants) | 117
  Abn E: Wk 30 (>=17 y) | 1.7
  Abn F: Wk 30 (>=17 y): number analyzed (Participants) | 117
  Abn F: Wk 30 (>=17 y) | 0.9
  Abn C: Wk 46 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn C: Wk 46 (>=12 y-<17 y) | 6.3
  Abn E: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn E: Wk 46 (>=17 y) | 1.2
  Abn B: Wk 62 (3 y-<12 y): number analyzed (Participants) | 10
  Abn B: Wk 62 (3 y-<12 y) | 20.0
  Abn C: Wk 62 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn C: Wk 62 (>=12 y-<17 y) | 6.3
  Abn E: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn E: Wk 62 (>=17 y) | 2.9
  Abn F: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn F: Wk 62 (>=17 y) | 0.6
  Abn E: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn E: Wk 78 (>=17 y) | 5.4
  Abn F: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn F: Wk 78 (>=17 y) | 1.8
  Abn G: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn G: Wk 78 (>=17 y) | 1.8
  Abn B: Wk 94 (3 y-<12 y): number analyzed (Participants) | 7
  Abn B: Wk 94 (3 y-<12 y) | 28.6
  Abn C: Wk 94 (>=12 y-<17 y): number analyzed (Participants) | 14
  Abn C: Wk 94 (>=12 y-<17 y) | 7.1
  Abn E: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn E: Wk 94 (>=17 y) | 2.7
  Abn F: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn F: Wk 94 (>=17 y) | 0.7
  Abn G: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn G: Wk 94 (>=17 y) | 0.7
  Abn D: Wk 118 (>=12 y-<17 y): number analyzed (Participants) | 2
  Abn D: Wk 118 (>=12 y-<17 y) | 50.0
  Abn E: Wk 142 (>=17 y): number analyzed (Participants) | 46
  Abn E: Wk 142 (>=17 y) | 8.7
  Abn F: Wk 142 (>=17 y): number analyzed (Participants) | 46
  Abn F: Wk 142 (>=17 y) | 2.2
  Abn E: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn E: Early TV (>=17 y) | 2.0
  Abn F: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn F: Early TV (>=17 y) | 2.0

43. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in 12-lead ECG Parameter (QRS Interval)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA ECG results of QRS interval were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '3 years -<12 years', the abnormality criteria were '>100 ms' (Abn A) and '>25% increase from Baseline' value (Abn B). For the age range, '>=12 years - <17 years', the abnormality criteria were '>110 ms' (Abn C) and '>25% increase from Baseline' (Abn D). For age range, '>=17 years', the abnormality criteria were treatment-emergent values above '>100 ms' (Abn E), '>120 ms' (Abn F), or '>140 ms' (Abn G).
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of ECG parameter (QRS interval) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Abn E: Wk 2 (>=17 y): number analyzed (Participants) | 196
  Abn E: Wk 2 (>=17 y) | 5.1
  Abn D: Wk 14 (>=12 y-<17 y): number analyzed (Participants) | 18
  Abn D: Wk 14 (>=12 y-<17 y) | 5.6
  Abn E: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn E: Wk 14 (>=17 y) | 9.9
  Abn F: Wk 14 (>=17 y): number analyzed (Participants) | 191
  Abn F: Wk 14 (>=17 y) | 0.5
  Abn E: Wk 30 (>=17 y): number analyzed (Participants) | 118
  Abn E: Wk 30 (>=17 y) | 7.6
  Abn A: Wk 46 (3 y-<12 y): number analyzed (Participants) | 12
  Abn A: Wk 46 (3 y-<12 y) | 8.3
  Abn D: Wk 46 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn D: Wk 46 (>=12 y-<17 y) | 6.3
  Abn E: Wk 46 (>=17 y): number analyzed (Participants) | 172
  Abn E: Wk 46 (>=17 y) | 7.6
  Abn D: Wk 62 (>=12 y-<17 y): number analyzed (Participants) | 16
  Abn D: Wk 62 (>=12 y-<17 y) | 6.3
  Abn E: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn E: Wk 62 (>=17 y) | 10.6
  Abn F: Wk 62 (>=17 y): number analyzed (Participants) | 170
  Abn F: Wk 62 (>=17 y) | 1.8
  Abn E: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn E: Wk 78 (>=17 y) | 8.9
  Abn F: Wk 78 (>=17 y): number analyzed (Participants) | 56
  Abn F: Wk 78 (>=17 y) | 1.8
  Abn C: Wk 94 (>=12 y-<17 y): number analyzed (Participants) | 14
  Abn C: Wk 94 (>=12 y-<17 y) | 7.1
  Abn D: Wk 94 (>=12 y-<17 y): number analyzed (Participants) | 14
  Abn D: Wk 94 (>=12 y-<17 y) | 7.1
  Abn E: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn E: Wk 94 (>=17 y) | 6.1
  Abn F: Wk 94 (>=17 y): number analyzed (Participants) | 148
  Abn F: Wk 94 (>=17 y) | 0.7
  Abn E: Wk 118 (>=17 y): number analyzed (Participants) | 21
  Abn E: Wk 118 (>=17 y) | 14.3
  Abn E: Wk 142 (>=17 y): number analyzed (Participants) | 47
  Abn E: Wk 142 (>=17 y) | 10.6
  Abn E: Early TV (>=17 y): number analyzed (Participants) | 49
  Abn E: Early TV (>=17 y) | 10.2
  Abn E: TV (>=17 y): number analyzed (Participants) | 36
  Abn E: TV (>=17 y) | 5.6
  Abn F: TV (>=17 y): number analyzed (Participants) | 36
  Abn F: TV (>=17 y) | 5.6

44. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in 12-lead ECG Parameter (Heart Rate Interval)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA ECG results of Heart rate interval were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '3 years -<12 years', the abnormality criteria were '<60 beats per minute (bpm)' (Abn A) and '>130 bpm' (Abn B). For the age range, '>=12 years', the abnormality criteria were '<50 bpm' (Abn C) and '>120 bpm' (Abn D).
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number of participants analyzed included those participants who were evaluable for the assessment. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of ECG parameter (Heart rate interval) observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 216
percentage of participants
  Abn C: Wk 2 (>=12 y) | 1.4
  Abn C: Wk 14 (>=12 y): number analyzed (Participants) | 209
  Abn C: Wk 14 (>=12 y) | 2.4
  Abn C: Wk 30 (>=12 y): number analyzed (Participants) | 130
  Abn C: Wk 30 (>=12 y) | 1.5
  Abn C: Wk 46 (>=12 y): number analyzed (Participants) | 188
  Abn C: Wk 46 (>=12 y) | 0.5
  Abn D: Wk 46 (>=12 y): number analyzed (Participants) | 188
  Abn D: Wk 46 (>=12 y) | 0.5
  Abn C: Wk 62 (>=12 y): number analyzed (Participants) | 186
  Abn C: Wk 62 (>=12 y) | 3.2
  Abn D: Wk 62 (>=12 y): number analyzed (Participants) | 186
  Abn D: Wk 62 (>=12 y) | 0.5
  Abn C: Wk 78 (>=12 y): number analyzed (Participants) | 61
  Abn C: Wk 78 (>=12 y) | 3.3
  Abn C: Wk 94 (>=12 y): number analyzed (Participants) | 162
  Abn C: Wk 94 (>=12 y) | 1.2
  Abn C: Wk 118 (>=12 y): number analyzed (Participants) | 23
  Abn C: Wk 118 (>=12 y) | 4.3
  Abn D: Wk 214 (>=12 y): number analyzed (Participants) | 1
  Abn D: Wk 214 (>=12 y) | 100
  Abn D: TV (>=12 y): number analyzed (Participants) | 43
  Abn D: TV (>=12 y) | 2.3

45. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Vital Sign Measurements (Pulse Rate)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA vital signs results of Pulse rate were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '3 years -<12 years', the abnormality criteria were '<60 bpm' (Low) and '>130 bpm' (High). For the age range, '12 years - <17 years', the abnormality criteria were '<=50 bpm' (Low) and '>=120 bpm' (High). For the age range, '>=17 years', the abnormality criteria were '<=50 bpm and a decrease from Baseline of >=15 bpm' (Low A), '>=120 bpm and an increase from Baseline of >=15 bpm' (High A), '<60 bpm' (Low B) and '>100 bpm' (High B). The Pulse rate was reported as per positions such as 'Supine 3 minute (Sup 3 min)', 'Standing 1 minute' (Std 1 min), and 'Standing 3 minute' (Std 3 min).
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Pulse rate observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Low B: Wk 2 (>=17 y)-Sup 3 min: number analyzed (Participants) | 199
  Low B: Wk 2 (>=17 y)-Sup 3 min | 4.5
  High B: Wk 2 (>=17 y)- Sup 3 min: number analyzed (Participants) | 199
  High B: Wk 2 (>=17 y)- Sup 3 min | 0.5
  High: Wk 2 (>=12 y-<17 y)-Std 1 min: number analyzed (Participants) | 20
  High: Wk 2 (>=12 y-<17 y)-Std 1 min | 5.0
  Low B: Wk 2 (>=17 y)-Std 1 min: number analyzed (Participants) | 197
  Low B: Wk 2 (>=17 y)-Std 1 min | 2.5
  High B: Wk 2 (>=17 y)-Std 1 min: number analyzed (Participants) | 197
  High B: Wk 2 (>=17 y)-Std 1 min | 3.0
  Low B: Wk 2 (>=17 y)-Std 3 min: number analyzed (Participants) | 196
  Low B: Wk 2 (>=17 y)-Std 3 min | 1.5
  High B: Wk 2 (>=17 y)-Std 3 min: number analyzed (Participants) | 196
  High B: Wk 2 (>=17 y)-Std 3 min | 2.6
  Low A: Wk 6 (>=17 y)-Sup 3 min: number analyzed (Participants) | 196
  Low A: Wk 6 (>=17 y)-Sup 3 min | 0.5
  Low B: Wk 6 (>=17 y)-Sup 3 min: number analyzed (Participants) | 196
  Low B: Wk 6 (>=17 y)-Sup 3 min | 4.6
  High B: Wk 6 (>=17 y)-Sup 3 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)-Sup 3 min | 2.0
  High: Wk 6 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 21
  High: Wk 6 (>=12 y-<17 y)- Std 1 min | 4.8
  Low B: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  Low B: Wk 6 (>=17 y)- Std 1 min | 1.5
  High B: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Std 1 min | 3.1
  Low A: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  Low A: Wk 6 (>=17 y)- Std 3 min | 0.5
  Low B: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  Low B: Wk 6 (>=17 y)- Std 3 min | 1.0
  High B: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Std 3 min | 2.6
  Low B: Wk 14 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  Low B: Wk 14 (>=17 y)- Sup 3 min | 4.1
  High B: Wk 14 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High B: Wk 14 (>=17 y)- Sup 3 min | 1.0
  High: Wk 14 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 18
  High: Wk 14 (>=12 y-<17 y)- Std 1 min | 5.6
  Low B: Wk 14 (>=17 y)- Std 1 min: number analyzed (Participants) | 195
  Low B: Wk 14 (>=17 y)- Std 1 min | 3.1
  High B: Wk 14 (>=17 y)- Std 1 min: number analyzed (Participants) | 195
  High B: Wk 14 (>=17 y)- Std 1 min | 2.6
  Low B: Wk 14 (>=17 y)- Std 3 min: number analyzed (Participants) | 195
  Low B: Wk 14 (>=17 y)- Std 3 min | 0.5
  High B: Wk 14 (>=17 y)- Std 3 min: number analyzed (Participants) | 195
  High B: Wk 14 (>=17 y)- Std 3 min | 4.1
  Low B: Wk 22 (>=17 y)- Sup 3 min: number analyzed (Participants) | 189
  Low B: Wk 22 (>=17 y)- Sup 3 min | 3.2
  High B: Wk 22 (>=17 y)- Sup 3 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Sup 3 min | 0.5
  High A: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  High A: Wk 22 (>=17 y)- Std 1 min | 0.5
  Low B: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  Low B: Wk 22 (>=17 y)- Std 1 min | 1.6
  High B: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Std 1 min | 4.2
  Low B: Wk 22 (>=17 y)- Std 3 min: number analyzed (Participants) | 189
  Low B: Wk 22 (>=17 y)- Std 3 min | 2.1
  High B: Wk 22 (>=17 y)- Std 3 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Std 3 min | 3.7
  Low B: Wk 30 (>=17 y)- Sup 3 min: number analyzed (Participants) | 119
  Low B: Wk 30 (>=17 y)- Sup 3 min | 1.7
  Low B: Wk 30 (>=17 y)- Std 1 min: number analyzed (Participants) | 119
  Low B: Wk 30 (>=17 y)- Std 1 min | 5.0
  High B: Wk 30 (>=17 y)- Std 1 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Std 1 min | 3.4
  Low B: Wk 30 (>=17 y)- Std 3 min: number analyzed (Participants) | 119
  Low B: Wk 30 (>=17 y)- Std 3 min | 2.5
  High B: Wk 30 (>=17 y)- Std 3 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Std 3 min | 1.7
  Low B: Wk 38 (>=17 y)- Sup 3 min: number analyzed (Participants) | 108
  Low B: Wk 38 (>=17 y)- Sup 3 min | 3.7
  Low B: Wk 38 (>=17 y)- Std 1 min: number analyzed (Participants) | 107
  Low B: Wk 38 (>=17 y)- Std 1 min | 2.8
  High B: Wk 38 (>=17 y)- Std 1 min: number analyzed (Participants) | 107
  High B: Wk 38 (>=17 y)- Std 1 min | 5.6
  Low B: Wk 38 (>=17 y)- Std 3 min: number analyzed (Participants) | 107
  Low B: Wk 38 (>=17 y)- Std 3 min | 0.9
  High B: Wk 38 (>=17 y)- Std 3 min: number analyzed (Participants) | 107
  High B: Wk 38 (>=17 y)- Std 3 min | 2.8
  Low B: Wk 46 (>=17 y)- Sup 3 min: number analyzed (Participants) | 174
  Low B: Wk 46 (>=17 y)- Sup 3 min | 5.7
  High B: Wk 46 (>=17 y)- Sup 3 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Sup 3 min | 1.7
  Low A: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  Low A: Wk 46 (>=17 y)- Std 1 min | 0.6
  High A: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  High A: Wk 46 (>=17 y)- Std 1 min | 1.1
  Low B: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  Low B: Wk 46 (>=17 y)- Std 1 min | 4.0
  High B: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Std 1 min | 5.2
  Low B: Wk 46 (>=17 y)- Std 3 min: number analyzed (Participants) | 174
  Low B: Wk 46 (>=17 y)- Std 3 min | 2.9
  High B: Wk 46 (>=17 y)- Std 3 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Std 3 min | 4.6
  Low B: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Sup 3 min | 5.2
  High B: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Sup 3 min | 2.3
  Low: Wk 62 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 16
  Low: Wk 62 (>=12 y-<17 y)- Std 1 min | 6.3
  High A: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  High A: Wk 62 (>=17 y)- Std 1 min | 0.6
  Low B: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Std 1 min | 4.6
  High B: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Std 1 min | 4.0
  High A: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  High A: Wk 62 (>=17 y)- Std 3 min | 0.6
  Low B: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Std 3 min | 2.3
  High B: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Std 3 min | 2.9
  Low B: Wk 78 (>=17 y)- Sup 3 min: number analyzed (Participants) | 60
  Low B: Wk 78 (>=17 y)- Sup 3 min | 6.7
  High B: Wk 78 (>=17 y)- Sup 3 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Sup 3 min | 1.7
  Low B: Wk 78 (>=17 y)- Std 1 min: number analyzed (Participants) | 60
  Low B: Wk 78 (>=17 y)- Std 1 min | 6.7
  High B: Wk 78 (>=17 y)- Std 1 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Std 1 min | 6.7
  Low B: Wk 78 (>=17 y)- Std 3 min: number analyzed (Participants) | 60
  Low B: Wk 78 (>=17 y)- Std 3 min | 6.7
  High B: Wk 78 (>=17 y)- Std 3 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Std 3 min | 5.0
  Low B: Wk 94 (>=17 y)- Sup 3 min: number analyzed (Participants) | 148
  Low B: Wk 94 (>=17 y)- Sup 3 min | 6.1
  High B: Wk 94 (>=17 y)- Sup 3 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Sup 3 min | 0.7
  Low B: Wk 94 (>=17 y)- Std 1 min: number analyzed (Participants) | 148
  Low B: Wk 94 (>=17 y)- Std 1 min | 2.7
  High B: Wk 94 (>=17 y)- Std 1 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Std 1 min | 4.1
  Low B: Wk 94 (>=17 y)- Std 3 min: number analyzed (Participants) | 148
  Low B: Wk 94 (>=17 y)- Std 3 min | 1.4
  High B: Wk 94 (>=17 y)- Std 3 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Std 3 min | 2.7
  Low B: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  Low B: Wk 118 (>=17 y)- Sup 3 min | 2.2
  High B: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  High B: Wk 118 (>=17 y)- Sup 3 min | 2.2
  Low B: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 90
  Low B: Wk 118 (>=17 y)- Std 1 min | 2.2
  High B: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 90
  High B: Wk 118 (>=17 y)- Std 1 min | 3.3
  Low B: Wk 118 (>=17 y)- Std 3 min: number analyzed (Participants) | 90
  Low B: Wk 118 (>=17 y)- Std 3 min | 2.2
  High B: Wk 118 (>=17 y)- Std 3 min: number analyzed (Participants) | 90
  High B: Wk 118 (>=17 y)- Std 3 min | 4.4
  High A: Wk 142 (>=17 y)- Sup 3 min: number analyzed (Participants) | 63
  High A: Wk 142 (>=17 y)- Sup 3 min | 1.6
  Low B: Wk 142 (>=17 y)- Sup 3 min: number analyzed (Participants) | 63
  Low B: Wk 142 (>=17 y)- Sup 3 min | 6.3
  High B: Wk 142 (>=17 y)- Sup 3 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Sup 3 min | 4.8
  High A: Wk 142 (>=17 y)- Std 1 min: number analyzed (Participants) | 63
  High A: Wk 142 (>=17 y)- Std 1 min | 3.2
  High B: Wk 142 (>=17 y)- Std 1 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Std 1 min | 7.9
  High A: Wk 142 (>=17 y)- Std 3 min: number analyzed (Participants) | 63
  High A: Wk 142 (>=17 y)- Std 3 min | 1.6
  Low B: Wk 142 (>=17 y)- Std 3 min: number analyzed (Participants) | 63
  Low B: Wk 142 (>=17 y)- Std 3 min | 3.2
  High B: Wk 142 (>=17 y)- Std 3 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Std 3 min | 7.9
  Low B: Wk 166 (>=17 y)- Sup 3 min: number analyzed (Participants) | 52
  Low B: Wk 166 (>=17 y)- Sup 3 min | 3.8
  High B: Wk 166 (>=17 y)- Sup 3 min: number analyzed (Participants) | 52
  High B: Wk 166 (>=17 y)- Sup 3 min | 1.9
  Low B: Wk 166 (>=17 y)- Std 1 min: number analyzed (Participants) | 51
  Low B: Wk 166 (>=17 y)- Std 1 min | 2.0
  High B: Wk 166 (>=17 y)- Std 1 min: number analyzed (Participants) | 51
  High B: Wk 166 (>=17 y)- Std 1 min | 5.9
  High B: Wk 166 (>=17 y)- Std 3 min: number analyzed (Participants) | 51
  High B: Wk 166 (>=17 y)- Std 3 min | 5.9
  Low B: Wk 190 (>=17 y)- Sup 3 min: number analyzed (Participants) | 34
  Low B: Wk 190 (>=17 y)- Sup 3 min | 2.9
  High B: Wk 190 (>=17 y)- Sup 3 min: number analyzed (Participants) | 34
  High B: Wk 190 (>=17 y)- Sup 3 min | 8.8
  High B: Wk 190 (>=17 y)- Std 1 min: number analyzed (Participants) | 34
  High B: Wk 190 (>=17 y)- Std 1 min | 11.8
  High B: Wk 190 (>=17 y)- Std 3 min: number analyzed (Participants) | 34
  High B: Wk 190 (>=17 y)- Std 3 min | 17.6
  High B: Wk 214 (>=17 y)- Sup 3 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Sup 3 min | 5.9
  High B: Wk 214 (>=17 y)- Std 1 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Std 1 min | 5.9
  High B: Wk 214 (>=17 y)- Std 3 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Std 3 min | 5.9
  Low B: Early TV (>=17 y)- Sup 3 min: number analyzed (Participants) | 55
  Low B: Early TV (>=17 y)- Sup 3 min | 3.6
  High B: Early TV (>=17 y)- Sup 3 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Sup 3 min | 1.8
  High: Early TV (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 3
  High: Early TV (>=12 y-<17 y)- Std 1 min | 33.3
  Low B: Early TV (>=17 y)- Std 1 min: number analyzed (Participants) | 55
  Low B: Early TV (>=17 y)- Std 1 min | 3.6
  High B: Early TV (>=17 y)- Std 1 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Std 1 min | 5.5
  Low A: TV (>=17 years)- Sup 3 min: number analyzed (Participants) | 50
  Low A: TV (>=17 years)- Sup 3 min | 2.0
  Low B: TV (>=17 years)- Sup 3 min: number analyzed (Participants) | 50
  Low B: TV (>=17 years)- Sup 3 min | 4.0
  High B: TV (>=17 years)- Sup 3 min: number analyzed (Participants) | 50
  High B: TV (>=17 years)- Sup 3 min | 2.0
  Low B: TV (>=17 years)- Std 1 min: number analyzed (Participants) | 50
  Low B: TV (>=17 years)- Std 1 min | 2.0
  High B: TV (>=17 years)- Std 1 min: number analyzed (Participants) | 50
  High B: TV (>=17 years)- Std 1 min | 4.0
  Low B: TV (>=17 years)- Std 3 min: number analyzed (Participants) | 50
  Low B: TV (>=17 years)- Std 3 min | 2.0
  High B: TV (>=17 years)- Std 3 min: number analyzed (Participants) | 50
  High B: TV (>=17 years)- Std 3 min | 2.0

46. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Vital Sign Measurements (Systolic Blood Pressure)
Description: TEMA values of Systolic Blood Pressure (BP) results were those that were observed post- BL during the Treatment Period but not present at Baseline. For the age range, '3 years -<12 years', the abnormality criteria were '<80 millimeters of mercury (mmHg)' (Low) and '>140 mmHg' (High). For the age range, '>=12 years - <17 years', the abnormality criteria were '<90 mmHg' (Low) and '>160 mmHg' (High). For the age range, '>=17 years', the abnormality criteria were '<=90 mmHg and decrease from Baseline of >=20 mmHg' (Low A), '>=180 mmHg and increase from Baseline of >=20' mmHg (High A), '<90 mmHg' (Low B), '>140 mmHg (High B), and '>160 mmHg' (High C). Systolic BP were reported as per positions such as 'Sup 3 min', 'Std 1 min, and 'Std 3 min'.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Systolic BP observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  High B: Wk 2 (>=17 y)- Sup 3 min: number analyzed (Participants) | 199
  High B: Wk 2 (>=17 y)- Sup 3 min | 3.5
  Low B: Wk 2 (>=17 y)- Std 1 min: number analyzed (Participants) | 197
  Low B: Wk 2 (>=17 y)- Std 1 min | 1.0
  High B: Wk 2 (>=17 y)- Std 1 min: number analyzed (Participants) | 197
  High B: Wk 2 (>=17 y)- Std 1 min | 2.5
  High B: Wk 2 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High B: Wk 2 (>=17 y)- Std 3 min | 3.6
  High B: Wk 6 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Sup 3 min | 3.1
  High B: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Std 1 min | 2.0
  Low B: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  Low B: Wk 6 (>=17 y)- Std 3 min | 0.5
  High B: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Std 3 min | 3.6
  Low B: Wk 14 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  Low B: Wk 14 (>=17 y)- Sup 3 min | 0.5
  High B: Wk 14 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High B: Wk 14 (>=17 y)- Sup 3 min | 3.1
  High B: Wk 14 (>=17 y)- Std 1 min: number analyzed (Participants) | 195
  High B: Wk 14 (>=17 y)- Std 1 min | 3.6
  High B: Wk 14 (>=17 y)- Std 3 min: number analyzed (Participants) | 195
  High B: Wk 14 (>=17 y)- Std 3 min | 3.6
  High B: Wk 22 (>=17 y)- Sup 3 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Sup 3 min | 4.2
  High B: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Std 1 min | 4.2
  High B: Wk 22 (>=17 y)- Std 3 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Std 3 min | 3.7
  Low B: Wk 30 (>=17 y)- Sup 3 min: number analyzed (Participants) | 119
  Low B: Wk 30 (>=17 y)- Sup 3 min | 0.8
  High B: Wk 30 (>=17 y)- Sup 3 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Sup 3 min | 5.9
  High B: Wk 30 (>=17 y)- Std 1 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Std 1 min | 2.5
  High B: Wk 30 (>=17 y)- Std 3 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Std 3 min | 5.0
  Low B: Wk 38 (>=17 y)- Sup 3 min: number analyzed (Participants) | 108
  Low B: Wk 38 (>=17 y)- Sup 3 min | 0.9
  High B: Wk 38 (>=17 y)- Sup 3 min: number analyzed (Participants) | 108
  High B: Wk 38 (>=17 y)- Sup 3 min | 2.8
  Low B: Wk 38 (>=17 y)- Std 1 min: number analyzed (Participants) | 107
  Low B: Wk 38 (>=17 y)- Std 1 min | 0.9
  High B: Wk 38 (>=17 y)- Std 1 min: number analyzed (Participants) | 107
  High B: Wk 38 (>=17 y)- Std 1 min | 2.8
  High B: Wk 38 (>=17 y)- Std 3 min: number analyzed (Participants) | 107
  High B: Wk 38 (>=17 y)- Std 3 min | 3.7
  Low: Wk 46 (>=12 y-<17 y)- Sup 3 min: number analyzed (Participants) | 16
  Low: Wk 46 (>=12 y-<17 y)- Sup 3 min | 6.3
  High B: Wk 46 (>=17 y)- Sup 3 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Sup 3 min | 2.9
  Low: Wk 46 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 16
  Low: Wk 46 (>=12 y-<17 y)- Std 1 min | 6.3
  High B: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Std 1 min | 2.3
  Low: Wk 46 (>=12 y-<17 y)- Std 3 min: number analyzed (Participants) | 16
  Low: Wk 46 (>=12 y-<17 y)- Std 3 min | 6.3
  High B: Wk 46 (>=17 y)- Std 3 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Std 3 min | 3.4
  High C: Wk 46 (>=17 y)- Std 3 min: number analyzed (Participants) | 174
  High C: Wk 46 (>=17 y)- Std 3 min | 0.6
  Low B: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Sup 3 min | 0.6
  High B: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Sup 3 min | 3.5
  Low: Wk 62 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 16
  Low: Wk 62 (>=12 y-<17 y)- Std 1 min | 6.3
  Low A: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  Low A: Wk 62 (>=17 y)- Std 1 min | 0.6
  Low B: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Std 1 min | 0.6
  High B: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Std 1 min | 2.3
  Low A: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  Low A: Wk 62 (>=17 y)- Std 3 min | 0.6
  Low B: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Std 3 min | 1.7
  High B: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Std 3 min | 1.2
  Low A: Wk 78 (>=17 y)- Sup 3 min: number analyzed (Participants) | 60
  Low A: Wk 78 (>=17 y)- Sup 3 min | 1.7
  High B: Wk 78 (>=17 y)- Sup 3 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Sup 3 min | 1.7
  High B: Wk 78 (>=17 y)- Std 1 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Std 1 min | 1.7
  High B: Wk 78 (>=17 y)- Std 3 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Std 3 min | 1.7
  High B: Wk 94 (>=17 y)- Sup 3 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Sup 3 min | 4.1
  High B: Wk 94 (>=17 y)- Std 1 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Std 1 min | 4.1
  High B: Wk 94 (>=17 y)- Std 3 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Std 3 min | 4.1
  High B: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  High B: Wk 118 (>=17 y)- Sup 3 min | 5.4
  High C: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  High C: Wk 118 (>=17 y)- Sup 3 min | 1.1
  High B: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 91
  High B: Wk 118 (>=17 y)- Std 1 min | 5.5
  High C: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 91
  High C: Wk 118 (>=17 y)- Std 1 min | 1.1
  High B: Wk 118 (>=17 y)- Std 3 min: number analyzed (Participants) | 91
  High B: Wk 118 (>=17 y)- Std 3 min | 6.6
  High C: Wk 118 (>=17 y)- Std 3 min: number analyzed (Participants) | 91
  High C: Wk 118 (>=17 y)- Std 3 min | 1.1
  High B: Wk 142 (>=17 y)- Sup 3 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Sup 3 min | 6.3
  High B: Wk 142 (>=17 y)- Std 1 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Std 1 min | 6.3
  High B: Wk 142 (>=17 y)- Std 3 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Std 3 min | 6.3
  High B: Wk 166 (>=17 y)- Sup 3 min: number analyzed (Participants) | 52
  High B: Wk 166 (>=17 y)- Sup 3 min | 3.8
  High B: Wk 166 (>=17 y)- Std 1 min: number analyzed (Participants) | 51
  High B: Wk 166 (>=17 y)- Std 1 min | 7.8
  High B: Wk 166 (>=17 y)- Std 3 min: number analyzed (Participants) | 51
  High B: Wk 166 (>=17 y)- Std 3 min | 7.8
  High B: Wk 190 (>=17 y)- Sup 3 min: number analyzed (Participants) | 34
  High B: Wk 190 (>=17 y)- Sup 3 min | 2.9
  High B: Wk 214 (>=17 y)- Std 1 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Std 1 min | 5.9
  High C: Wk 214 (>=17 y)- Std 1 min: number analyzed (Participants) | 17
  High C: Wk 214 (>=17 y)- Std 1 min | 5.9
  High B: Wk 214 (>=17 y)- Std 3 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Std 3 min | 5.9
  High B: Wk 262 (>=17 y)- Std 3 min: number analyzed (Participants) | 1
  High B: Wk 262 (>=17 y)- Std 3 min | 100
  High B: Early TV (>=17 y)- Sup 3 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Sup 3 min | 1.8
  High B: Early TV (>=17 y)- Std 1 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Std 1 min | 1.8
  High B: TV (>=17 y)- Std 1 min: number analyzed (Participants) | 50
  High B: TV (>=17 y)- Std 1 min | 4.0
  High B: TV (>=17 y)- Std 3 min: number analyzed (Participants) | 50
  High B: TV (>=17 y)- Std 3 min | 2.0

47. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Vital Sign Measurements (Diastolic Blood Pressure)
Description: TEMA values of Diastolic BP results were those that are observed post- BL during the Treatment Period but not present at Baseline. For the age range, '3 years -<12 years', the abnormality criteria were '<50 mmHg' (Low) and '>80 mmHg' (High), '>=12 years - <17 years', the abnormality criteria were '<=50 mmHg' (Low) and '>=105 mmHg' (High), and '>=17 years', the abnormality criteria were '<=50 mmHg and decrease from Baseline of >=15 mmHg' (Low A), '>=105 mmHg and increase from Baseline of >=15' mmHg (High A), '<50 mmHg' (Low B), '>90 mmHg' (High B), and '>100 mmHg' (High C). Diastolic BP were reported as per positions such as 'Sup 3 min', 'Std 1 min, and 'Std 3 min'.
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA value of Diastolic BP observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  Low: Wk 2 (3 y-<12 y)- Sup 3 min: number analyzed (Participants) | 16
  Low: Wk 2 (3 y-<12 y)- Sup 3 min | 6.3
  Low B: Wk 2 (>=17 y)- Sup 3 min: number analyzed (Participants) | 199
  Low B: Wk 2 (>=17 y)- Sup 3 min | 0.5
  High B: Wk 2 (>=17 y)- Sup 3 min: number analyzed (Participants) | 199
  High B: Wk 2 (>=17 y)- Sup 3 min | 2.5
  Low: Wk 2 (3 y-<12 y)- Std 1 min: number analyzed (Participants) | 16
  Low: Wk 2 (3 y-<12 y)- Std 1 min | 6.3
  High: Wk 2 (3 y-<12 y)- Std 1 min: number analyzed (Participants) | 16
  High: Wk 2 (3 y-<12 y)- Std 1 min | 6.3
  High B: Wk 2 (>=17 y)- Std 1 min: number analyzed (Participants) | 197
  High B: Wk 2 (>=17 y)- Std 1 min | 5.1
  High C: Wk 2 (>=17 y)- Std 1 min: number analyzed (Participants) | 197
  High C: Wk 2 (>=17 y)- Std 1 min | 0.5
  Low: Wk 2 (3 y-<12 y)- Std 3 min: number analyzed (Participants) | 16
  Low: Wk 2 (3 y-<12 y)- Std 3 min | 6.3
  High: Wk 2 (3 y-<12 y)- Std 3 min: number analyzed (Participants) | 16
  High: Wk 2 (3 y-<12 y)- Std 3 min | 12.5
  High B: Wk 2 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High B: Wk 2 (>=17 y)- Std 3 min | 6.1
  High C: Wk 2 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High C: Wk 2 (>=17 y)- Std 3 min | 0.5
  Low A: Wk 6 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  Low A: Wk 6 (>=17 y)- Sup 3 min | 0.5
  High B: Wk 6 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Sup 3 min | 4.6
  High C: Wk 6 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High C: Wk 6 (>=17 y)- Sup 3 min | 0.5
  Low A: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  Low A: Wk 6 (>=17 y)- Std 1 min | 0.5
  High A: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  High A: Wk 6 (>=17 y)- Std 1 min | 0.5
  High B: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Std 1 min | 4.1
  High C: Wk 6 (>=17 y)- Std 1 min: number analyzed (Participants) | 196
  High C: Wk 6 (>=17 y)- Std 1 min | 0.5
  High: Wk 6 (3 y-<12 y)- Std 3 min: number analyzed (Participants) | 14
  High: Wk 6 (3 y-<12 y)- Std 3 min | 7.1
  Low A: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  Low A: Wk 6 (>=17 y)- Std 3 min | 0.5
  Low B: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  Low B: Wk 6 (>=17 y)- Std 3 min | 0.5
  High B: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High B: Wk 6 (>=17 y)- Std 3 min | 6.6
  High C: Wk 6 (>=17 y)- Std 3 min: number analyzed (Participants) | 196
  High C: Wk 6 (>=17 y)- Std 3 min | 0.5
  High: Wk 14 (3 y-<12 y)- Sup 3 min: number analyzed (Participants) | 13
  High: Wk 14 (3 y-<12 y)- Sup 3 min | 7.7
  High B: Wk 14 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High B: Wk 14 (>=17 y)- Sup 3 min | 2.0
  High C: Wk 14 (>=17 y)- Sup 3 min: number analyzed (Participants) | 196
  High C: Wk 14 (>=17 y)- Sup 3 min | 0.5
  High A: Wk 14 (>=17 y)- Std 1 min: number analyzed (Participants) | 195
  High A: Wk 14 (>=17 y)- Std 1 min | 0.5
  High B: Wk 14 (>=17 y)- Std 1 min: number analyzed (Participants) | 195
  High B: Wk 14 (>=17 y)- Std 1 min | 3.1
  High C: Wk 14 (>=17 y)- Std 1 min: number analyzed (Participants) | 195
  High C: Wk 14 (>=17 y)- Std 1 min | 1.0
  High: Wk 14 (3 y-<12 y)- Std 3 min: number analyzed (Participants) | 12
  High: Wk 14 (3 y-<12 y)- Std 3 min | 8.3
  High B: Wk 14 (>=17 y)- Std 3 min: number analyzed (Participants) | 195
  High B: Wk 14 (>=17 y)- Std 3 min | 4.6
  High C: Wk 14 (>=17 y)- Std 3 min: number analyzed (Participants) | 195
  High C: Wk 14 (>=17 y)- Std 3 min | 0.5
  High: Wk 22 (3 y-<12 y)- Sup 3 min: number analyzed (Participants) | 13
  High: Wk 22 (3 y-<12 y)- Sup 3 min | 15.4
  Low: Wk 22 (>=12 y-<17 y)- Sup 3 min: number analyzed (Participants) | 16
  Low: Wk 22 (>=12 y-<17 y)- Sup 3 min | 6.3
  High B: Wk 22 (>=17 y)- Sup 3 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Sup 3 min | 1.6
  High C: Wk 22 (>=17 y)- Sup 3 min: number analyzed (Participants) | 189
  High C: Wk 22 (>=17 y)- Sup 3 min | 0.5
  High: Wk 22 (3 y-<12 y)- Std 1 min: number analyzed (Participants) | 13
  High: Wk 22 (3 y-<12 y)- Std 1 min | 15.4
  Low A: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  Low A: Wk 22 (>=17 y)- Std 1 min | 1.1
  Low B: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  Low B: Wk 22 (>=17 y)- Std 1 min | 0.5
  High B: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Std 1 min | 7.9
  High C: Wk 22 (>=17 y)- Std 1 min: number analyzed (Participants) | 189
  High C: Wk 22 (>=17 y)- Std 1 min | 0.5
  High: Wk 22 (3 y-<12 y)- Std 3 min: number analyzed (Participants) | 13
  High: Wk 22 (3 y-<12 y)- Std 3 min | 7.7
  Low A: Wk 22 (>=17 y)- Std 3 min: number analyzed (Participants) | 189
  Low A: Wk 22 (>=17 y)- Std 3 min | 0.5
  High B: Wk 22 (>=17 y)- Std 3 min: number analyzed (Participants) | 189
  High B: Wk 22 (>=17 y)- Std 3 min | 6.3
  High C: Wk 22 (>=17 y)- Std 3 min: number analyzed (Participants) | 189
  High C: Wk 22 (>=17 y)- Std 3 min | 1.1
  High B: Wk 30 (>=17 y)- Sup 3 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Sup 3 min | 3.4
  High C: Wk 30 (>=17 y)- Sup 3 min: number analyzed (Participants) | 119
  High C: Wk 30 (>=17 y)- Sup 3 min | 0.8
  High: Wk 30 (3 y-<12 y)- Std 1 min: number analyzed (Participants) | 7
  High: Wk 30 (3 y-<12 y)- Std 1 min | 14.3
  High A: Wk 30 (>=17 y)- Std 1 min: number analyzed (Participants) | 119
  High A: Wk 30 (>=17 y)- Std 1 min | 0.8
  High B: Wk 30 (>=17 y)- Std 1 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Std 1 min | 5.9
  High C: Wk 30 (>=17 y)- Std 1 min: number analyzed (Participants) | 119
  High C: Wk 30 (>=17 y)- Std 1 min | 0.8
  High B: Wk 30 (>=17 y)- Std 3 min: number analyzed (Participants) | 119
  High B: Wk 30 (>=17 y)- Std 3 min | 4.2
  High B: Wk 38 (>=17 y)- Sup 3 min: number analyzed (Participants) | 108
  High B: Wk 38 (>=17 y)- Sup 3 min | 2.8
  High: Wk 38 (3 y-<12 y)- Std 1 min: number analyzed (Participants) | 5
  High: Wk 38 (3 y-<12 y)- Std 1 min | 20.0
  High B: Wk 38 (>=17 y)- Std 1 min: number analyzed (Participants) | 107
  High B: Wk 38 (>=17 y)- Std 1 min | 5.6
  High C: Wk 38 (>=17 y)- Std 1 min: number analyzed (Participants) | 107
  High C: Wk 38 (>=17 y)- Std 1 min | 0.9
  High B: Wk 38 (>=17 y)- Std 3 min: number analyzed (Participants) | 107
  High B: Wk 38 (>=17 y)- Std 3 min | 9.3
  Low A: Wk 46 (>=17 y)- Sup 3 min: number analyzed (Participants) | 174
  Low A: Wk 46 (>=17 y)- Sup 3 min | 0.6
  High B: Wk 46 (>=17 y)- Sup 3 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Sup 3 min | 4.0
  Low: Wk 46 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 16
  Low: Wk 46 (>=12 y-<17 y)- Std 1 min | 6.3
  High B: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Std 1 min | 8.0
  High C: Wk 46 (>=17 y)- Std 1 min: number analyzed (Participants) | 174
  High C: Wk 46 (>=17 y)- Std 1 min | 0.6
  High B: Wk 46 (>=17 y)- Std 3 min: number analyzed (Participants) | 174
  High B: Wk 46 (>=17 y)- Std 3 min | 9.8
  High C: Wk 46 (>=17 y)- Std 3 min: number analyzed (Participants) | 174
  High C: Wk 46 (>=17 y)- Std 3 min | 1.1
  High A: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  High A: Wk 62 (>=17 y)- Sup 3 min | 0.6
  High B: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Sup 3 min | 5.2
  High C: Wk 62 (>=17 y)- Sup 3 min: number analyzed (Participants) | 173
  High C: Wk 62 (>=17 y)- Sup 3 min | 1.2
  High: Wk 62 (3 y-<12 y)- Std 1 min: number analyzed (Participants) | 10
  High: Wk 62 (3 y-<12 y)- Std 1 min | 20.0
  Low: Wk 62 (>=12 y-<17 y)- Std 1 min: number analyzed (Participants) | 16
  Low: Wk 62 (>=12 y-<17 y)- Std 1 min | 6.3
  High A: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  High A: Wk 62 (>=17 y)- Std 1 min | 0.6
  High B: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Std 1 min | 5.8
  High C: Wk 62 (>=17 y)- Std 1 min: number analyzed (Participants) | 173
  High C: Wk 62 (>=17 y)- Std 1 min | 1.2
  Low B: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  Low B: Wk 62 (>=17 y)- Std 3 min | 0.6
  High B: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  High B: Wk 62 (>=17 y)- Std 3 min | 5.8
  High C: Wk 62 (>=17 y)- Std 3 min: number analyzed (Participants) | 173
  High C: Wk 62 (>=17 y)- Std 3 min | 0.6
  Low: Wk 78 (>=12 y-<17 y)- Sup 3 min: number analyzed (Participants) | 6
  Low: Wk 78 (>=12 y-<17 y)- Sup 3 min | 16.7
  High B: Wk 78 (>=17 y)- Sup 3 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Sup 3 min | 1.7
  High B: Wk 78 (>=17 y)- Std 1 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Std 1 min | 3.3
  High B: Wk 78 (>=17 y)- Std 3 min: number analyzed (Participants) | 60
  High B: Wk 78 (>=17 y)- Std 3 min | 3.3
  High C: Wk 78 (>=17 y)- Std 3 min: number analyzed (Participants) | 60
  High C: Wk 78 (>=17 y)- Std 3 min | 1.7
  High B: Wk 94 (>=17 y)- Sup 3 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Sup 3 min | 1.4
  High B: Wk 94 (>=17 y)- Std 1 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Std 1 min | 4.1
  High: Wk 94 (3 y-<12 y)- Std 3 min: number analyzed (Participants) | 7
  High: Wk 94 (3 y-<12 y)- Std 3 min | 14.3
  High A: Wk 94 (>=17 y)- Std 3 min: number analyzed (Participants) | 148
  High A: Wk 94 (>=17 y)- Std 3 min | 0.7
  High B: Wk 94 (>=17 y)- Std 3 min: number analyzed (Participants) | 148
  High B: Wk 94 (>=17 y)- Std 3 min | 4.7
  High C: Wk 94 (>=17 y)- Std 3 min: number analyzed (Participants) | 148
  High C: Wk 94 (>=17 y)- Std 3 min | 0.7
  Low A: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  Low A: Wk 118 (>=17 y)- Sup 3 min | 1.1
  High A: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  High A: Wk 118 (>=17 y)- Sup 3 min | 1.1
  Low B: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  Low B: Wk 118 (>=17 y)- Sup 3 min | 1.1
  High B: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  High B: Wk 118 (>=17 y)- Sup 3 min | 2.2
  High C: Wk 118 (>=17 y)- Sup 3 min: number analyzed (Participants) | 92
  High C: Wk 118 (>=17 y)- Sup 3 min | 1.1
  Low A: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 91
  Low A: Wk 118 (>=17 y)- Std 1 min | 1.1
  Low B: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 91
  Low B: Wk 118 (>=17 y)- Std 1 min | 1.1
  High B: Wk 118 (>=17 y)- Std 1 min: number analyzed (Participants) | 91
  High B: Wk 118 (>=17 y)- Std 1 min | 4.4
  High B: Wk 118 (>=17 y)- Std 3 min: number analyzed (Participants) | 91
  High B: Wk 118 (>=17 y)- Std 3 min | 7.7
  High B: Wk 142 (>=17 y)- Sup 3 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Sup 3 min | 6.3
  High B: Wk 142 (>=17 y)- Std 1 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Std 1 min | 7.9
  High B: Wk 142 (>=17 y)- Std 3 min: number analyzed (Participants) | 63
  High B: Wk 142 (>=17 y)- Std 3 min | 7.9
  High B: Wk 166 (>=17 y)- Sup 3 min: number analyzed (Participants) | 52
  High B: Wk 166 (>=17 y)- Sup 3 min | 3.8
  High B: Wk 166 (>=17 y)- Std 1 min: number analyzed (Participants) | 51
  High B: Wk 166 (>=17 y)- Std 1 min | 5.9
  High A: Wk 166 (>=17 y)- Std 3 min: number analyzed (Participants) | 51
  High A: Wk 166 (>=17 y)- Std 3 min | 2.0
  High B: Wk 166 (>=17 y)- Std 3 min: number analyzed (Participants) | 51
  High B: Wk 166 (>=17 y)- Std 3 min | 11.8
  High C: Wk 166 (>=17 y)- Std 3 min: number analyzed (Participants) | 51
  High C: Wk 166 (>=17 y)- Std 3 min | 2.0
  High B: Wk 190 (>=17 y)- Std 3 min: number analyzed (Participants) | 34
  High B: Wk 190 (>=17 y)- Std 3 min | 2.9
  High B: Wk 214 (>=17 y)- Sup 3 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Sup 3 min | 5.9
  High A: Wk 214 (>=17 y)- Std 1 min: number analyzed (Participants) | 17
  High A: Wk 214 (>=17 y)- Std 1 min | 5.9
  High B: Wk 214 (>=17 y)- Std 1 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Std 1 min | 5.9
  High C: Wk 214 (>=17 y)- Std 1 min: number analyzed (Participants) | 17
  High C: Wk 214 (>=17 y)- Std 1 min | 5.9
  High A: Wk 214 (>=17 y)- Std 3 min: number analyzed (Participants) | 17
  High A: Wk 214 (>=17 y)- Std 3 min | 5.9
  High B: Wk 214 (>=17 y)- Std 3 min: number analyzed (Participants) | 17
  High B: Wk 214 (>=17 y)- Std 3 min | 5.9
  High C: Wk 214 (>=17 y)- Std 3 min: number analyzed (Participants) | 17
  High C: Wk 214 (>=17 y)- Std 3 min | 5.9
  High B: Early TV (>=17 y)- Sup 3 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Sup 3 min | 3.6
  High C: Early TV (>=17 y)- Sup 3 min: number analyzed (Participants) | 55
  High C: Early TV (>=17 y)- Sup 3 min | 1.8
  High B: Early TV (>=17 y)- Std 1 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Std 1 min | 9.1
  High C: Early TV (>=17 y)- Std 1 min: number analyzed (Participants) | 55
  High C: Early TV (>=17 y)- Std 1 min | 1.8
  High A: Early TV (>=17 y)- Std 3 min: number analyzed (Participants) | 55
  High A: Early TV (>=17 y)- Std 3 min | 1.8
  High B: Early TV (>=17 y)- Std 3 min: number analyzed (Participants) | 55
  High B: Early TV (>=17 y)- Std 3 min | 10.9
  High C: Early TV (>=17 y)- Std 3 min: number analyzed (Participants) | 55
  High C: Early TV (>=17 y)- Std 3 min | 3.6
  High: TV (3 y-<12 y)- Sup 3 min: number analyzed (Participants) | 6
  High: TV (3 y-<12 y)- Sup 3 min | 16.7
  High B: TV (>=17 y)- Sup 3 min: number analyzed (Participants) | 50
  High B: TV (>=17 y)- Sup 3 min | 4.0
  High B: TV (>=17 y)- Std 1 min: number analyzed (Participants) | 50
  High B: TV (>=17 y)- Std 1 min | 2.0
  High B: TV (>=17 y)- Std 3 min: number analyzed (Participants) | 50
  High B: TV (>=17 y)- Std 3 min | 4.0
  High C: TV (>=17 y)- Std 3 min: number analyzed (Participants) | 50
  High C: TV (>=17 y)- Std 3 min | 2.0

48. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Marked Abnormalities (TEMAs) in Vital Sign Measurements (Body Weight)
Description: TEMA values are defined in the SAP as significant deviations from the expected range of age-appropriate values. TEMA vital signs parameter results were those that are observed post- BL during the Treatment Period but not present at Baseline. For the age range, '1 month - <17 years', the abnormality criteria were '<3% of normal body weight' in Kilograms (kg) or '>97% of normal body weight' in kgs. Here, '<3% of normal' is presented as 'Low' and '>97% of normal' is presented as 'High'. For the age range '>=17 years', the abnormality criteria were 'Increase/decrease of >=10%' body weight in kgs (presented as Inc/Dec A) or 'Increase/decrease of >=7%' body weight in kgs (presented as Inc/Dec B).
Time Frame: During the study (up to approximately 5 years)
Population: The Safety Set included all study participants who received at least 1 dose of IMP during this study. Number analyzed signifies participants who were evaluable at specified time points. Data for visits wherein at least 1 TEMA body weight value observed during the study were reported in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 239
percentage of participants
  High- Wk 14 (1 m - <17 y): number analyzed (Participants) | 31
  High- Wk 14 (1 m - <17 y) | 9.7
  Inc/Dec A- Wk 14 (>=17 y): number analyzed (Participants) | 195
  Inc/Dec A- Wk 14 (>=17 y) | 5.6
  Inc/Dec B- Wk 14 (>=17 y): number analyzed (Participants) | 195
  Inc/Dec B- Wk 14 (>=17 y) | 16.4
  High- Wk 30 (1 m - <17 y): number analyzed (Participants) | 19
  High- Wk 30 (1 m - <17 y) | 10.5
  Inc/Dec A- Wk 30 (>=17 y): number analyzed (Participants) | 119
  Inc/Dec A- Wk 30 (>=17 y) | 5.9
  Inc/Dec B- Wk 30 (>=17 y): number analyzed (Participants) | 119
  Inc/Dec B- Wk 30 (>=17 y) | 19.3
  High- Wk 46 (1 m - <17 y): number analyzed (Participants) | 28
  High- Wk 46 (1 m - <17 y) | 7.1
  Inc/Dec A- Wk 46 (>=17 y): number analyzed (Participants) | 177
  Inc/Dec A- Wk 46 (>=17 y) | 12.4
  Inc/Dec B- Wk 46 (>=17 y): number analyzed (Participants) | 177
  Inc/Dec B- Wk 46 (>=17 y) | 22.6
  High- Wk 62 (1 m - <17 y): number analyzed (Participants) | 26
  High- Wk 62 (1 m - <17 y) | 7.7
  Inc/Dec A- Wk 62 (>=17 y): number analyzed (Participants) | 174
  Inc/Dec A- Wk 62 (>=17 y) | 14.9
  Inc/Dec B- Wk 62 (>=17 y): number analyzed (Participants) | 174
  Inc/Dec B- Wk 62 (>=17 y) | 21.8
  Inc/Dec A- Wk 78 (>=17 y): number analyzed (Participants) | 63
  Inc/Dec A- Wk 78 (>=17 y) | 19.0
  Inc/Dec B- Wk 78 (>=17 y): number analyzed (Participants) | 63
  Inc/Dec B- Wk 78 (>=17 y) | 30.2
  High- Wk 94 (1 m - <17 y): number analyzed (Participants) | 23
  High- Wk 94 (1 m - <17 y) | 13.0
  Inc/Dec A- Wk 94 (>=17 y): number analyzed (Participants) | 152
  Inc/Dec A- Wk 94 (>=17 y) | 16.4
  Inc/Dec B- Wk 94 (>=17 y): number analyzed (Participants) | 152
  Inc/Dec B- Wk 94 (>=17 y) | 30.9
  Low- Wk 118 (1 m - <17 y): number analyzed (Participants) | 19
  Low- Wk 118 (1 m - <17 y) | 5.3
  High- Wk 118 (1 m - <17 y): number analyzed (Participants) | 19
  High- Wk 118 (1 m - <17 y) | 10.5
  Inc/Dec A- Wk 118 (>=17 y): number analyzed (Participants) | 97
  Inc/Dec A- Wk 118 (>=17 y) | 21.6
  Inc/Dec B- Wk 118 (>=17 y): number analyzed (Participants) | 97
  Inc/Dec B- Wk 118 (>=17 y) | 33.0
  Low- Wk 142 (1 m - <17 y): number analyzed (Participants) | 13
  Low- Wk 142 (1 m - <17 y) | 7.7
  High- Wk 142 (1 m - <17 y): number analyzed (Participants) | 13
  High- Wk 142 (1 m - <17 y) | 7.7
  Inc/Dec A- Wk 142 (>=17 y): number analyzed (Participants) | 77
  Inc/Dec A- Wk 142 (>=17 y) | 19.5
  Inc/Dec B- Wk 142 (>=17 y): number analyzed (Participants) | 77
  Inc/Dec B- Wk 142 (>=17 y) | 32.5
  High- Wk 166 (1 m - <17 y): number analyzed (Participants) | 10
  High- Wk 166 (1 m - <17 y) | 10.0
  Inc/Dec A- Wk 166 (>=17 y): number analyzed (Participants) | 60
  Inc/Dec A- Wk 166 (>=17 y) | 25.0
  Inc/Dec B- Wk 166 (>=17 y): number analyzed (Participants) | 60
  Inc/Dec B- Wk 166 (>=17 y) | 45.0
  Low- Wk 190 (1 m - <17 y): number analyzed (Participants) | 6
  Low- Wk 190 (1 m - <17 y) | 16.7
  Inc/Dec A- Wk 190 (>=17 y): number analyzed (Participants) | 46
  Inc/Dec A- Wk 190 (>=17 y) | 26.1
  Inc/Dec B- Wk 190 (>=17 y): number analyzed (Participants) | 46
  Inc/Dec B- Wk 190 (>=17 y) | 50.0
  Low- Wk 214 (1 m - <17 y): number analyzed (Participants) | 2
  Low- Wk 214 (1 m - <17 y) | 50.0
  Inc/Dec A- Wk 214 (>=17 y): number analyzed (Participants) | 22
  Inc/Dec A- Wk 214 (>=17 y) | 31.8
  Inc/Dec B- Wk 214 (>=17 y): number analyzed (Participants) | 22
  Inc/Dec B- Wk 214 (>=17 y) | 54.5
  Inc/Dec A- Wk 238 (>=17 y): number analyzed (Participants) | 6
  Inc/Dec A- Wk 238 (>=17 y) | 16.7
  Inc/Dec B- Wk 238 (>=17 y): number analyzed (Participants) | 6
  Inc/Dec B- Wk 238 (>=17 y) | 50.0
  Inc/Dec A- Wk 262 (>=17 y): number analyzed (Participants) | 3
  Inc/Dec A- Wk 262 (>=17 y) | 33.3
  Inc/Dec B- Wk 262 (>=17 y): number analyzed (Participants) | 3
  Inc/Dec B- Wk 262 (>=17 y) | 33.3
  Inc/Dec A- Early TV (>=17 y): number analyzed (Participants) | 57
  Inc/Dec A- Early TV (>=17 y) | 26.3
  Inc/Dec B- Early TV (>=17 y): number analyzed (Participants) | 57
  Inc/Dec B- Early TV (>=17 y) | 33.3
  High- TV (1 m - <17 y): number analyzed (Participants) | 14
  High- TV (1 m - <17 y) | 21.4
  Inc/Dec A- TV (>=17 y): number analyzed (Participants) | 55
  Inc/Dec A- TV (>=17 y) | 34.5
  Inc/Dec B- TV (>=17 y): number analyzed (Participants) | 55
  Inc/Dec B- TV (>=17 y) | 52.7

49. Secondary Outcome: Percent Change in Primary Generalized Tonic-clonic Seizure (PGTCS) Frequency Per 28 Days From Combined Baseline
Description: The 28-day PGTCS frequency during the relative period was subtracted from the 28-day Combined Baseline PGTCS frequency and the result was divided by 28-day Combined Baseline PGTCS frequency and the result was then multiplied by 100 to get percent change in PGTCS frequency per 28 days from Combined Baseline Period (CB) to the appropriate analysis Period. The CB was defined as the combined 12-week Historical Baseline and 4-week Prospective Baseline periods immediately prior to randomization in the study SP0982 or prior to Visit 1 (first dose) if direct enrollers in EP0012.
Time Frame: From Combined Baseline until end of Treatment Period (up to approximately 5 years)
Population: Full Analysis Set (FAS) was a subset of the Safety Set and included all study participants with seizure diary data for at least 1 day during this study.
Measure: Median (Full Range); unit: percent change
Arm/Group | All Participants (Lacosamide)
Number analyzed (Participants) | 238
percent change | -88.58 [-100.0 to 465.4]

ADVERSE EVENTS:
Time Frame: From Visit 1 (Week 0) to End of Treatment Period (up to approximately 5 years)
Description: AEs were considered treatment-emergent if event had onset on or after date of first study medication dose in EP0012 and within 30 days following last study medication dose or events whose intensity worsened on or after date of first study medication dose and within 30 days following date of last study medication administration. TEAEs were assessed on SS.
Arm/Group | All Participants (Lacosamide)
All-Cause Mortality (participants affected / at risk) | 4/239
Serious Adverse Events (participants affected / at risk) | 54/239
Other Adverse Events (participants affected / at risk) | 176/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (Lacosamide) (N=239)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Drowning (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (4)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Periorbital contusion (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Drug level increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 16 (20)
Status epilepticus (Nervous system disorders) | 4 (7)
Myoclonic epilepsy (Nervous system disorders) | 2 (2)
Petit mal epilepsy (Nervous system disorders) | 1 (2)
Benign intracranial hypertension (Nervous system disorders) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Psychogenic seizure (Psychiatric disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (Lacosamide) (N=239)
Vertigo (Ear and labyrinth disorders) | 19 (30)
Diplopia (Eye disorders) | 12 (15)
Nausea (Gastrointestinal disorders) | 23 (31)
Diarrhoea (Gastrointestinal disorders) | 18 (23)
Vomiting (Gastrointestinal disorders) | 16 (24)
Fatigue (General disorders) | 13 (15)
Pyrexia (General disorders) | 13 (13)
Nasopharyngitis (Infections and infestations) | 52 (91)
Influenza (Infections and infestations) | 18 (23)
Upper respiratory tract infection (Infections and infestations) | 17 (18)
Corona virus infection (Infections and infestations) | 14 (16)
Contusion (Injury, poisoning and procedural complications) | 24 (30)
Laceration (Injury, poisoning and procedural complications) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (19)
Headache (Nervous system disorders) | 56 (113)
Dizziness (Nervous system disorders) | 53 (73)
Somnolence (Nervous system disorders) | 40 (51)
Grand mal convulsion (Nervous system disorders) | 14 (16)
Migraine (Nervous system disorders) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02408549/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02408549/SAP_001.pdf